

# STATISTICAL ANALYSIS PLAN

Study CRO-PK-20-344 - Sponsor code Z7251J01

# Comparative bioavailability study of a new riluzole orodispersible film vs. a marketed oral reference (Rilutek® tablets) in healthy male and female volunteers

Single centre, single dose, open-label, randomised, 2-sequence, 4-period replicate cross-over study

Test formulation: Riluzole 50 mg orodispersible film, Aquestive Therapeutics, USA

Reference formulation: Rilutek®, 50 mg riluzole tablets, Sanofi Mature IP, France

Sponsor: Zambon S.p.A., via Lillo del Duca 10, I-20091 Bresso, Italy

Phone: +39.02.66.52.42.99 Fax: +39.02.66.52.48.87

Email: carlo.cattaneo@zambongroup.com

Investigator: Milko Radicioni, MD - Principal investigator

CROSS Research S.A., Phase I Unit

Via F.A. Giorgioli 14

CH-6864 Arzo, Switzerland Phone: +41.91.64.04.450 Fax: +41.91.64.04.451

Email: clinic@croalliance.com

Development phase: I

Version and date: Final version 1.0, 31MAY2021

This study will be conducted in accordance with current version of Good Clinical Practice (GCP), ICH topic E6 (R2)

Property of the sponsor
May not be used, divulged, published or otherwise disclosed without the consent of the sponsor

This document comprises 33 pages plus appendices



# **VERSIONS' HISTORY**

| Version | Date of Issue | Reason for change |
|---|---|---|
| Draft version 0.1 | 21MAY2021 | Alice Segantin issued the first draft |
| Draft version 0.2 | 28MAY2021 | Alice Segantin issued the second draft after revision of MW |
| Final version 1.0 | 31MAY2021 | Alice Segantin issued the final version after sponsor approval |



# APPROVAL AND ACKNOWLEDGEMENT

**SPONSOR** 

Zambon S.p.A., Italy

Sponsor Representative (for approval and acknowledgement)

Carlo Cattaneo, Global Head Medical Affairs CNS

Date

Signature





| CRO | |
|---|---|
| CROSS Research S.A. | |
| Biometry Unit Representative<br>Alessandra Gentili, Biometry M | (for approval and acknowledgement) [anager, Unit Head] |
| 31MAY2021 | Aforerefel! |
| Date | Signature |
| Statistical Analysis (for appro | |
| Alice Segantin, Clinical program | |
| BAMAY 2021 | Alice feautin |
| Date | Signature |
| Medical Writing | |
| Andrea Di Stefano, Senior Med | ical Writer and PK Expert |
| OZJUNZOZŁ | andread Style |
| Date | Signature |
| Coordination (for acknowledge Elena Gander, Clinical Project I | |
| 011. [000] | Samo Clauder |

Signature



# STUDY/INVESTIGATION SCHEDULE

| ACTIVITIES | Screening | PERIOD 1. 2 | 3 4 (wash-c | out>7 days) | Final<br>visit/ETV <sup>12</sup> |
|---|---|---|---|---|---|
| Visit | V1 | V2, V4, V6, V8 | PERIOD 1, 2, 3, 4 (wash-out≥7 days)<br>V2, V4, V6, V8 V3, V5, V7, V9 | | V10 <sup>11</sup> /ETV |
| , 1910 | Days -14/-2 | Day -1 | Day 1 | Day 2 | Day 2 <sup>11</sup> /ETV |
| Informed consent | X | • | • | • | |
| Demography | Х | | | | |
| Lifestyle | X | | | | |
| Medical/surgical history | X | | | | |
| Physical abnormalities | X | | | | X |
| Previous and concomitant treatments | x | X | X | X | X |
| Height | Х | | | | |
| Body weight | Х | | | | X |
| Laboratory analysis <sup>1</sup> | Х | | | | X |
| Cotinine | Х | | | | |
| Virology | Х | | | | |
| Drug screening | X | X | | | |
| Vital signs | X | | x <sup>2</sup> | x <sup>2</sup> | x <sup>13</sup> |
| Pregnancy test | x <sup>3</sup> | x <sup>4</sup> | | | |
| ECG | X | | | | |
| Inclusion/exclusion criteria | X | x <sup>5</sup> | | | |
| Eligibility evaluation | X | x <sup>5</sup> | | | |
| Alcohol breath test | | X | | | |
| Enrolment and randomisation | | x <sup>5</sup> | | | |
| Confinement | | X | X | | |
| Discharge | | | | X | |
| IMP administration | | | x <sup>6</sup> | | |
| Palatability | | | x <sup>7</sup> | | |
| Mouth visual inspection | | | x <sup>8</sup> | | |
| Blood samplings <sup>9</sup> | | | X | X | |
| Standardised meals | | X | X | X | |
| AEs monitoring <sup>10</sup> | X | X | X | X | X |

- 1. Haematology, blood chemistry with the exception of cotinine, urinalysis
- 2. At pre-dose and 2 and 36 h post-dose
- 3. Women only serum  $\beta$ -HCG test
- 4. Women only urine test
- 5. Period 1, visit 2
- 6. At  $08:00 \pm 1$  h under fasting conditions
- 7. Immediately after each administration of the test product
- 8. At pre-dose and 0.5 and 1 h post-dose at each administration of the test product
- 9. At pre-dose (0) and 15, 30, 45 min, 1, 1.25, 1.5, 2, 3, 4, 6, 8, 12, 24 and 36 h post-dose
- 10. Adverse events monitored starting at the screening visit, immediately after informed consent, up to the final visit/ETV
- 11. Final visit on Day 2 of period 4 after the 36-h post-dose blood sampling
- 12. Early termination visit (ETV) in case of subject's premature discontinuation
- 13. At the ETV only



# TABLES OF CONTENTS

| | STATISTICAL ANALYSIS PLAN | 1 |
|---|---|---|
| | VERSIONS' HISTORY | 2 |
| | APPROVAL AND ACKNOWLEDGEMENT | 3 |
| | STUDY/INVESTIGATION SCHEDULE | 5 |
| | TABLES OF CONTENTS | 6 |
| | TABLES | 7 |
| | ABBREVIATIONS | 8 |
| 1 | INTRODUCTION | 10 |
| 1.1 | Changes with respect to the study protocol and its amendment | 10 |
| 2 | STUDY OBJECTIVES | 11 |
| 2.1 | Primary end-point | 11 |
| 2.2 | Secondary end-points | 11 |
| 3 | INVESTIGATIONAL PLAN | 12 |
| 3.1 | Overall study design | 12 |
| 3.2 | Discussion of design | 12 |
| 4 | STUDY POPULATION | 13 |
| 4.1 | Target population | 13 |
| 4.2 | Inclusion criteria | 13 |
| 4.3 | Exclusion criteria | 13 |
| 4.3.1 | Not allowed treatments | 14 |
| 5 | STUDY SCHEDULE | 16 |
| 5.1 | Study visits and procedures | 16 |
| 5.2 | Diet and lifestyle | 19 |
| 5.3 | Restrictions | 19 |
| 6 | STUDY SUBJECT IDENTIFICATION METHOD AND TREATMENT ASSIGNMENT METHOD | 20 |
| 6.1 | Unique subject identifier | 20 |
| <b>6.2</b> | Subject identifier for the study | 20 |
| 6.3 | Randomisation | 20 |
| 6.4 | Treatment allocation | 20 |
| 6.5 | Blinding | 20 |
| 7 | STUDY EVALUATION PARAMETERS | 21 |
| 7.1 | Study variables | 21 |
| 7.1.1 | Primary variables | 21 |
| 7.1.2 | Secondary variables | 21 |
| 7.2 | Pharmacokinetic assessments | 21 |
| 7.2.1 | Pharmacokinetic parameters | 21 |
| 7.3 | Safety and tolerability parameters | 22 |
| 8 | STATISTICAL METHOD | 23 |
| 8.1 | Tables, listings and figures layout | 23 |
| 8.2 | <b>Analysis sets</b> | 24 |
| 8.2.1 | Definitions | 24 |
| 8.2.1.1 | Reasons for exclusion from the PK Set before bioanalysis | 24 |
| 8.2.1.2 | Reasons for exclusion from the PK Set after bioanalysis | 25 |
| 8.3 | Sample size and power considerations | 25 |





| 8.4 | Demographic, baseline and background characteristics | 26 |
|---|---|---|
| 8.4.1 | Subjects' disposition | 26 |
| 8.4.2 | <b>Analysis sets</b> | 26 |
| 8.4.3 | | |
| 8.4.4 | B.4.4 Discontinued subjects | |
| 8.4.5 | Protocol deviations | 26 |
| 8.4.6 | Demography | 27 |
| 8.4.7 | Inclusion/exclusion criteria not met | 27 |
| 8.4.8 | ECG | 27 |
| 8.4.9 | Medical and surgical history | 27 |
| 8.4.10 | Prior and concomitant medication | 27 |
| 8.4.11 | Subjects' study visits | 27 |
| 8.4.12 | Fertility status and contraceptive method | 27 |
| 8.4.13 | Alcohol breath test, pregnancy test, cotinine test and urine drug test | 27 |
| 8.4.14 | Tobacco consumption | 28 |
| 8.4.15 | Meals | 28 |
| 8.5 | IMP administration | 28 |
| 8.5.1 | Dose per body weight | 28 |
| 8.5.2 | Wash-out | 28 |
| 8.6 | PK and Palatability analysis | 28 |
| 8.6.1 | PK blood samples collection | 28 |
| 8.6.2 | Descriptive pharmacokinetics/pharmacodynamics | 28 |
| 8.6.3 | Statistical comparison of pharmacokinetic parameters | 29 |
| <b>8.7</b> | Safety and tolerability analysis | 30 |
| 8.7.1 | Adverse events | 30 |
| 8.7.2 | Vital signs | 31 |
| 8.7.3 | Laboratory data | 31 |
| 8.7.4 | Physical examination | 31 |
| 8.7.5 | Mouth Visual Inspection | 31 |
| 8.8 | Analysis datasets | 31 |
| 9 | REFERENCES | 32 |
| 10 | APPENDICES | 33 |
| | TABLES | |
| Table 9.4 | .1 - Sample size calculation | 25 |
| Table 8.9 actual CV | | 30 |



# **ABBREVIATIONS**

AE Adverse Event

ANOVA Analysis of Variance

AUC<sub>0-t</sub> Area under the concentration-time curve from time zero to time t AUC<sub>0- $\infty$ </sub> Area under the concentration versus time curve up to infinity

%AUCextra Percentage of the residual area extrapolated to infinity in relation to the AUC∞

BE Bioequivalence

BLQL Below Lower Quantification Limit

BMI Body Mass Index BP Blood Pressure bpm Beats per minute BW Body weight

CDISC Clinical Data Interchange Standards Consortium

CI Confidence Interval

C<sub>max</sub> Peak drug concentration

CPL Clinical Project Leader

CRF Case Report Form

CRO Contract Research Organisation

CSP Clinical Study Protocol
CRS Clinical Study Report
CS Clinically Significant
CV Coefficient of Variation

CV<sub>WR</sub> Coefficient of Variation within-subject

DIABP Diastolic Blood Pressure

EC Ethics Committee ECG Electrocardiogram

EMA European Medicine Agency ETV Early Termination Visit

FDA Food and Drug Administration

FSFV First Subject First Visit GCP Good Clinical Practice GLP Good Laboratory Practice

HR Heart Rate

ICH International Conference on Harmonisation

IMP Investigational Medicinal Product

IUD Intra-Uterine Device

 $\lambda_z$  Terminal elimination rate constant, calculated, if feasible, by log-linear

regression using at least 3 points

LSLV Last Subject Last Visit

MedDRA Medical Dictionary for Regulatory Activities

min Minute N Normal

NA Not Applicable NC Not calculated

NCS Not clinically significant

OTC Over The Counter
PK Pharmacokinetics
PT Preferred Term





PTAE Pre-Treatment Adverse Event

QTc Corrected QT interval

R Reference

SAE Serious Adverse Event
SYSBP Systolic Blood Pressure
SD Standard Deviation
SOC System Organ Class

SOP Standard Operating Procedure SDTM Study Data Tabulation Model

SUSAR Suspected Unexpected Serious Adverse Reaction

T Test

TEAE Treatment-Emergent Adverse Event

 $t_{1/2}$  Half-life

t<sub>max</sub> Time to achieve Cmax

USDA United States Department of Agriculture

WHODDE World Health Organisation Drug Dictionary Enhanced



#### 1 INTRODUCTION

Statistical analysis will be performed by the CROSS Research Biometry Unit. The end-points and methods of analysis specified in this SAP are consistent with ICH E6 (R2) and E9 guidelines (1, 2) and with EMA guideline on the investigation of bioequivalence (3, 4). The SAP has been compiled by the CRO Biometry Unit on the basis of the final version 1.0 of the clinical study protocol and its amendment (5, 6), reviewed by the Sponsor and finalized before the database lock.

# 1.1 Changes with respect to the study protocol and its amendment

No change with respect to the study protocol and its amendment (5, 6) was introduced in this SAP.



# 2 STUDY OBJECTIVES

The objective of the study is to compare the pharmacokinetic profile of riluzole after replicate single dose of the novel orodispersible film test formulation and of the marketed reference Rilutek® tablets and to evaluate their bioequivalence.

# 2.1 Primary end-point

• To evaluate the bioequivalent rate  $(C_{max})$  and extent  $(AUC_{0-t})$  of absorption of riluzole after replicate single dose administration of test and reference.

# 2.2 Secondary end-points

- To describe the PK profile of riluzole after replicate single dose administration of test and reference;
- to evaluate the test product palatability;
- to collect safety and tolerability data of test and reference after replicate single dose administration.

CROSS Research S.A. Page 11



#### 3 INVESTIGATIONAL PLAN

# 3.1 Overall study design

Single centre, single dose, open-label, randomised, 2-sequence, 4-period replicate cross-over study.

# 3.2 Discussion of design

The study was designed in agreement with the EMA guideline "Guidance on the investigation of bioequivalence", CPMP/EWP/QWP/1401/98 Rev. 1 January 2010 (3). The well-known high variability of riluzole led to the choice of the replicate cross-over design as suggested by the current EMA guideline. According to the guideline, an enlargement of the acceptance interval for bioequivalence in terms of  $C_{max}$  is allowed up to 69.84-143.19% in relation to the actual intra-subject variability of riluzole  $C_{max}$  found in this study with the reference treatment, by keeping in consideration the favourable safety profile of the test formulation previously observed in 3 clinical studies. In detail, a  $C_{max}$  within-subject variability >30% was found in the previous pilot study and =32.66% in the previous bioequivalence study performed in USA (7). According to the 2-arm cross-over study design, each randomised subject will be allocated to one of 2 sequences of IMP administrations in the 4 study periods according to a computer generated randomisation list (see § 6.3). Balance between the sequences will be made so that subjects have the same chances to be assigned to either sequence (either RTRT or TRTR in the 4 consecutive periods).

An open-label design will be used since the primary end-point of the study is based on objective measurements of riluzole in plasma and the outcome variables could not be influenced by the subjects or investigator being aware of the administered products. The bioanalysis will be performed under blinded conditions.

The washout period of 7 days was estimated to be adequate. Based upon a half-life of 12 h (Rilutek SmPC reference: 8), it is anticipated that minimal plasma levels would be achieved in 5 days thus allowing dosing every 7 days. Blood sampling time-points were selected on the basis of the known PK profile of riluzole and on the basis of previous Phase I studies of the same test formulation administered to healthy volunteers.

The dose for the present study was selected based on EMA Rilutek<sup>®</sup> European Public Assessment Report (EPAR) (9), which recommends a dose regimen of 50 mg (one filmcoated tablet) twice a day in the common clinical practice. The dose of 50 mg is the minimal unit dose.



#### 4 STUDY POPULATION

# 4.1 Target population

Healthy men and women will be enrolled in this study.

#### 4.2 Inclusion criteria

To be enrolled in this study, subjects must fulfil all these criteria:

- 1. *Informed consent:* signed written informed consent before inclusion in the study
- 2. Sex and Age: men/women, 18-55 years old inclusive
- 3. *Tobacco:* non-smokers for at least 6 months prior to study screening
- 4. Body Mass Index (BMI): 18.5-29 kg/m2 inclusive
- 5. *Vital signs: systolic* blood pressure (SBP) 100-139 mmHg, diastolic blood pressure (DBP) 50-89 mmHg, heart rate 50-90 bpm, measured after 5 min at rest in the sitting position
- 6. Full comprehension: ability to comprehend the full nature and purpose of the study,
- 7. including possible risks and side effects; ability to co-operate with the investigator and to comply with the requirements of the entire study
- 8. *Contraception and fertility (women only):* women of child-bearing potential must be using at least one of the following reliable methods of contraception:
  - a. A non-hormonal intrauterine device [IUD] or female condom with spermicide or contraceptive sponge with spermicide or diaphragm with spermicide or cervical cap with spermicide for at least 2 months before the screening visit
  - b. A male sexual partner who agrees to use a male condom with spermicide
  - c. A sterile sexual partner

Female participants of non-child-bearing potential or in post-menopausal status for at least 1 year will be admitted.

For all women, pregnancy test result must be negative at screening.

#### 4.3 Exclusion criteria

Subjects meeting any of these criteria will not be enrolled in the study:

- 1. Electrocardiogram (ECG) 12-leads: (supine position) clinically significant abnormalities; QTc interval > 450 msec
- 2. *Physical findings:* clinically significant abnormal physical findings which could interfere with the objectives of the study
- 3. Laboratory analyses: clinically significant abnormal laboratory values indicative of physical illness
- 4. Cotinine: positive cotinine test at screening



- 5. Allergy: ascertained or presumptive hypersensitivity to the active principle and/or formulations' ingredients; history of anaphylaxis to drugs or allergic reactions in general, which the investigator considers may affect the outcome of the study
- 6. Diseases: clinically significant history or presence of renal, hepatic, gastrointestinal, cardiovascular, cerebrovascular, immunological, musculoskeletal, respiratory, skin, haematological, endocrine, psychiatric or neurological diseases or surgeries that may interfere with the aim of the study. Gastrointestinal pathologies include any clinically significant disorder of the mouth, e.g. impairment of swallowing, lesions, ulcerations, deformities, untreated dental caries
- 7. *Dentures:* presence of mouth jewellery, dentures, braces, piercings that may interfere with successful completion of the dosing
- 8. *Medications:* medications, including over the counter (OTC) medications and herbal remedies for 2 weeks before study screening; central nervous system depressants, including opioids, benzodiazepines, general anaesthetics and anticonvulsants, or CYP inhibitors, including cimetidine, fluoxetine, quinidine, erythromycin, ciprofloxacin, fluconazole, ketoconazole, diltiazem and antiretroviral agents, or strong CYP inducers, including barbiturates, carbamazepine, glucocorticoids, phenytoin, St John's wort and rifampin, or hormonal oral or transdermal contraceptives for 30 days before study screening; implanted, injected, intravaginal or intrauterine hormonal contraceptives for 6 months before study screening
- 9. *Investigative drug studies*: participation in the evaluation of any investigational product for 3 months before this study. The 3-month interval is calculated as the time between the first calendar day of the month that follows the last visit of the previous study and the first day of the present study
- 10. Blood donation: blood donations for 3 months before this study
- 11. Drug, alcohol, caffeine, tobacco: history of drug, alcohol [>1 drink/day for females and >2 drinks/day for males, defined according to the USDA Dietary Guidelines 2015 (10)], caffeine (>5 cups coffee/tea/day) or tobacco use including any tobacco product like ecigarettes and vaping products
- 12. Drug test: positive result at the drug test at screening or Day -1
- 13. Alcohol test: positive alcohol breath test at Day -1
- 14. Diet: abnormal diets (<1600 or >3500 kcal/day) or substantial changes in eating habits in the 4 weeks before this study; vegetarians and vegans
- 15. Pregnancy (women only): positive or missing pregnancy test at screening or Day -1, pregnant or lactating women

#### 4.3.1 Not allowed treatments

No medication, including OTC and herbal remedies, will be allowed for 2 weeks before the start of the study and during the whole study duration.

Central nervous system depressants, including opioids, benzodiazepines, general anaesthetics and anticonvulsants, or CYP inhibitors, including cimetidine, fluoxetine, quinidine, erythromycin, ciprofloxacin, fluconazole, ketoconazole, diltiazem and antiretroviral agents, or strong CYP inducers, including barbiturates, carbamazepine, glucocorticoids, phenytoin, St John's wort and rifampin, or hormonal oral or transdermal contraceptives will be forbidden for 30 days before study screening and during the whole study duration.

Implanted, injected, intravaginal or intrauterine hormonal contraceptives will be forbidden for





6 months before study screening and during the whole study duration.

Paracetamol will be allowed as therapeutic counter-measure for adverse events (AEs) according to the investigator's opinion.

The intake of any other medication will be reported as a protocol deviation. However, it will lead to subject's discontinuation from the study only if the investigator, together with the sponsor, considers it could affect the study assessments or outcome



#### 5 STUDY SCHEDULE

The schedule of the study/investigation is summarised at page 5.

# 5.1 Study visits and procedures

Each study subject will undergo 10 visits.

The study protocol foresees 4 periods separated by wash-out intervals of at least 7 days. Minimum study duration will be 25 days, screening visit included. A written informed consent will be obtained before any study assessment or procedure.

The first subject first visit (FSFV) is defined as the 1st visit performed at the Phase I Unit by the 1st screened subject. The last subject last visit (LSLV) is defined as the last visit performed at the Phase I Unit by the last subject, i.e. the last visit foreseen by the study protocol, independently of the fact that the subject is a completer or a withdrawn subject, and it corresponds to the study completion.

The following phases, visits and procedures will be performed:

- Screening phase
  - Screening visit 1: between Day -14 and Day -2
  - Period 1 visit 2: Day -1
- Interventional phase
  - Period 1 visit 3: Days 1-2
  - Wash-out interval of at least 7 days
  - ➤ Period 2 visit 4: Day -1
  - Period 2 visit 5: Days 1-2
  - Wash-out interval of at least 7 days
  - Period 3 visit 6: Day -1
  - Period 3 visit 7: Days 1-2
  - ➤ Wash-out interval of at least 7 days
  - ➤ Period 4 visit 8: Day -1
  - Period 4 visit 9: Days 1-2
- Final phase
  - ➤ Period 4 visit 10: Day 2 Final visit or early termination visit (ETV) in case of early discontinuation



| | | Day | Procedures/Assessments | Notes |
|---|---|---|---|---|
| Screening phase | Screening – visit 1 | From Day -14 to<br>Day -2 | <ul> <li>Explanation to the subject of study aims, procedures and possible risks</li> <li>Informed consent signature</li> <li>Screening number (as S001, S002, etc.)</li> <li>Demographic data and life style recording</li> <li>Medical/surgical history</li> <li>Previous/concomitant medications</li> <li>Full physical examination (body weight, height, vital signs, physical abnormalities)</li> <li>ECG recording</li> <li>Laboratory analyses: haematology, blood chemistry, cotinine, urinalysis, virology and serum pregnancy test (women only)</li> <li>Urine multi-drug kit test</li> <li>AE monitoring</li> <li>Inclusion/exclusion criteria evaluation</li> <li>Eligibility evaluation</li> </ul> | Note: The first two letters of the surname followed by the first two letters of the first name will be used in the Phase I Unit source document only and will not be transferred to the sponsor |
| | Visit 2 | Day -1 | <ul> <li>Alcohol breath test</li> <li>Urine multi-drug kit test</li> <li>Urine pregnancy test (women only)</li> <li>AE and concomitant medications</li> <li>Inclusion/exclusion criteria evaluation</li> <li>Eligibility evaluation</li> <li>Enrolment and randomisation</li> </ul> | Arrival at the Phase I Unit in the evening Confinement until the evening of Day 2 Standardised low-fat dinner Fasting for at least 10 h (overnight) up to dosing |
| Period 1 | | | <ul> <li>IMP administration at 08:00 ± 1 h</li> <li>Palatability of the test product immediately after administration</li> <li>Mouth visual inspections after administration of the test investigational medicinal product, at pre-dose and 0.5 and 1 h post-dose</li> <li>Vital signs measurement</li> <li>Blood sample collection for PK analysis</li> <li>AE and concomitant medications</li> </ul> | Fasting until about 5<br>h post-dose<br>Standardised lunch at<br>about 13:00<br>Standardised dinner<br>at about 20:00 (12 h<br>post-dose) |
| | Visit 3 | Day 2 | <ul> <li>Vital signs measurement</li> <li>Blood sample collection for PK analysis</li> <li>AE and concomitant medications</li> </ul> | Standardised breakfast at about 8:00 and lunch at about 13:00 Discharge from the Phase I Unit in the evening after the 36-h post-dose blood sample collection and vital signs check |
| At least 7 days At least 7 days A wash-out interval of at least 7 do consecutive administrations | | A wash-out interval of at least 7 days between 2 consecutive administrations | | |



| | | Day | Procedures/Assessments | Notes |
|---|---|---|---|---|
| 2 | Visit 4 | Day -1 | As visit 2, excluding inclusion/exclusion criteria evaluation, enrolment and randomisation | As visit 2 |
| Period 2 | Visit 5 | Day I | As visit 3. Test or reference IMP administered according to the randomisation list and cross-over design | As visit 3 |
| | Vis | Day 2 | As visit 3 | As visit 3 |
| West, est | w asn-out | At least 7 days | A wash-out interval of at least 7 days between 2 consecutive administrations | |
| | Visit 6 | Day -1 | As visit 2, excluding inclusion/exclusion criteria evaluation, enrolment and randomisation | As visit 2 |
| Period 3 | Visit 7 | Day I | As visit 3. Test or reference IMP administered according to the randomisation list and cross-over design | As visit 3 |
| | Vis | Day 2 | As visit 3 | As visit 3 |
| | | At least 7 days | A wash-out interval of at least 7 days between 2 consecutive administrations | |
| As visit 2, excluding inclusion/exclusion criteria evaluation, enrolment and randomisation | | As visit 2 | | |
| Period 4 | Visit 9 | Day 1 | As visit 3. Test or reference IMP administered according to the randomisation list and cross-over design | As visit 3 |
| Period 4 | Visit 9 | Day 2 | As visit 3 As visit 3 | |



| | | Day | Procedures/Assessments | Notes |
|---|---|---|---|---|
| Final phase | Visit 10 - Final Visit or ETV | Day 2 of<br>period 4 /<br>at ETV in case<br>of<br>discontinuation | <ul> <li>Full physical examination (body weight and physical abnormalities; also vital signs in case of ETV)</li> <li>Laboratory analyses as at screening, with the exception of cotinine, virology, urine drug test and pregnancy test</li> <li>AE and concomitant medications</li> <li>In case of clinically significant results at the final visit, the subjects will be followed-up by the investigator until the normalisation of the concerned clinical parameter(s)</li> </ul> | Upon leaving, the subjects will be instructed to contact immediately the investigator in case of occurrence of any adverse reactions |

# 5.2 Diet and lifestyle

During confinement, the subjects will not take any food or drinks (except water) for about 10 h (i.e. overnight) before IMP administration and for about 5 h afterwards. On Day -1 of each study period, a standardised low-fat dinner will be served. Water will be allowed as desired, except for one h before and one h after IMP administration. In order to maintain an adequate hydration, the subjects will be encouraged to drink at least 150 mL of still mineral water every 2 h for 5 h post-dose, starting at 1 h post-dose.

On Day 1 of each study period, the subjects will remain fasted until about 5 h post-dose. Standardised lunch and dinner will be served at approximately 5 h and 12 h post-dose. On Day 2 of each study period, standardised breakfast and lunch will be served at about 8:00 and 13:00, respectively. The meals' composition will be standardised on Days -1 and 1 in each study period (see the study protocol (5) for further details).

Coffee, tea or food containing xanthines (i.e. coke, chocolate, etc.), smoking, alcohol and grapefruit will be forbidden during confinement. In particular, alcohol and grapefruit will be forbidden for 24 h before the first IMP administration until the end of the study.

Only non-smokers will be included in the study.

During confinement, routine ambulant daily activities will be strongly recommended.

#### 5.3 Restrictions

During each study period, the subjects will be confined from the evening preceding the IMP administration (study Day -1) until the evening of Day 2.

For the 4 h following each administration, when not involved in study activities, the subjects will remain seated. They will not be allowed to lie down.

During confinement, hazardous, strenuous or athletic activities will not be permitted.



# 6 STUDY SUBJECT IDENTIFICATION METHOD AND TREATMENT ASSIGNMENT METHOD

# 6.1 Unique subject identifier

All the subjects who sign the informed consent form for the present study will be coded with "unique subject identifiers" when data are extracted from the study database into the domains of the CDISC SDTM and ADaM models. The unique subject identifier consists of the sponsor study code (i.e. Z7251J01), the 3-digit centre number (e.g. 001, 002, etc.), the 4-digit screening number (e.g. S001, S002, etc.) and the 3-digit randomisation number (e.g. 001, 002, etc., when applicable). Study code, centre number, screening number and randomisation number (when applicable) are separated by slashes ("/").

# 6.2 Subject identifier for the study

The last 8 digits of the unique subject identifier (enrolled subjects), corresponding to the subject screening and subject randomisation numbers separated by a slash, or the last 4 digits of the unique subject identifier (not enrolled subjects), corresponding to the subject screening number, will appear as subject identifier in the individual listings and figures of the clinical study report and will be used to identify the subjects in in-text tables or wording (if applicable).

# 6.3 Randomisation

The randomisation list was computer-generated by the Biometry Unit of the Clinical Contract Research Organization (CRO), using the PLAN procedure of the SAS® version 9.3 (TS1M1) (11). The randomisation list was supplied to the study site and to STM Pharma PRO Srl., Italy for the preparation of the IMP individual kits before study start and will be attached to the final clinical study report.

#### 6.4 Treatment allocation

The study subjects will be assigned to one of 2 sequences of treatments (either RTRT or TRTR) according to their randomisation number. Randomisation number will be given to the subjects on study Day -1, period 1, as soon as they are definitely enrolled in the study.

# 6.5 Blinding

This is an open study. No masking procedure will be applied.



#### 7 STUDY EVALUATION PARAMETERS

# 7.1 Study variables

# 7.1.1 Primary variables

• C<sub>max</sub> and AUC<sub>0-t</sub> of plasma riluzole after replicate single dose administration of test and reference formulation.

# 7.1.2 Secondary variables

- AUC<sub>0- $\infty$ </sub>,  $t_{1/2}$ ,  $t_{max}$ , AUC<sub>extra</sub>,  $\lambda_z$ , of riluzole after replicate single dose administration of test and reference;
- Palatability score
- TEAEs, vital signs (BP, HR), laboratory parameters, physical examination including BW

# 7.2 Pharmacokinetic assessments

The following PK parameters will be measured and/or calculated for riluzole, using the validated software Phoenix WinNonlin<sup>®</sup> version 6.3 (12) or higher (actual version will be stated in the final report).

# 7.2.1 Pharmacokinetic parameters

| • | $C_{max}$ | Maximum plasma concentration |
|---|---|---|
| • | $t_{max}$ | Time to achieve C <sub>max</sub> |
| • | $\lambda_{ m z}$ | Terminal elimination rate constant, calculated, if feasible, by log- |
| | | linear regression using at least 3 points |
| • | $t_{1/2}$ | Half-life, calculated, if feasible, as $ln(2)/\lambda_z$ |
| • | $\mathrm{AUC}_{0\text{-t}}$ | Area under the concentration-time curve from administration to the last observed concentration time t, calculated with the linear trapezoidal method |
| • | $AUC_{0\text{-}\infty}$ | Area under the concentration-time curve extrapolated to infinity, calculated, if feasible, as $AUC_{0-t} + C_t/\lambda_z$ , where $C_t$ is the last measurable drug concentration |
| • | %AUCextra | Percentage of the residual area $(C_t/\lambda_z)$ extrapolated to infinity in relation to the total $AUC_{0-\infty}$ , calculated, if feasible, as $100\times[(C_t/\lambda_z)/AUC_{0-\infty}]$ |

The sampling schedule is considered adequate if the ratio  $AUC_{0-t}/AUC_{0-\infty}$  equals or exceeds a factor of 0.8 (i.e. if %AUC<sub>extra</sub> is <20%) for more than 80% of the individual PK profiles. This assures that the primary variable AUC<sub>0-t</sub> covers a sufficient percentage of the theoretical total extent of exposure.

The quality of log-linear regression (and, consequently, the reliability of the extrapolated PK parameters) should be demonstrated by a determination coefficient  $R_2 \ge 0.8$ . Individual extrapolated parameters, when considered unreliable, will be reported as NC (not calculated).





# 7.3 Safety and tolerability parameters

Safety and general tolerability of the IMP will be based on TEAEs, physical examinations including body weight, vital signs and routine haematology, blood chemistry and urinalysis laboratory tests.



#### 8 STATISTICAL METHOD

The statistical analysis of demographic and safety data will be performed using SAS® version 9.3 (TS1M1) (11) or higher (the actual versions will be stated in the final report).

The statistical analysis of PK parameters will be performed using Phoenix WinNonlin<sup>®</sup> version 6.3 (12) or higher and SAS<sup>®</sup> version 9.3 (TS1M1) or higher.

The data documented in this study and the parameters measured will be evaluated and compared using classic descriptive statistics, i.e. geometric mean (PK data only), arithmetic mean, SD, CV (%), minimum, median and maximum values for quantitative variables and frequencies for qualitative variables.

# 8.1 Tables, listings and figures layout

Tables, listings and figures will be provided according to the following settings:

- Background: White
- Foreground: Black
- Font face: Times
- Font style: Roman
- Font size: 10 pt
- Font weight: Medium (data, footers and notes), Bold (titles and headers)
- Font width: Normal
- Layout: Landscape
- Top Margin: 2.5 cm
- Bottom Margin: 2.5 cm
- Left Margin: 0.8 cm
- Right Margin: 0.8 cm
- Test label: Riluzole 50 mg orodispersible film (T)
- Reference/Placebo label: Rilutek<sup>®</sup>, 50 mg riluzole tablets (R)
- Date format: ddMMMyyyy
- Means, standard deviations, percent coefficient of variations, medians, lower confidence limits and upper confidence limits will be rounded to one digit more than the original data
- Minima and maxima will keep the same number of decimal digits as the source values
- p-values will be rounded to the fourth decimal digit and will be flagged by an asterisk (\*) in case of statistical significance (i.e. p-value < 0.05 or, in case of centre by treatment interaction, p-value < 0.10)
- p-values lower than 0.0001 will be reported as "<.0001 \*".

The data and results of Riluzole 50 mg orodispersible film (T) will be presented before the data and results of Rilutek<sup>®</sup>, 50 mg riluzole tablets (R) in all listings and tables.



# 8.2 Analysis sets

#### 8.2.1 Definitions

A subject will be defined as <u>screened</u> after the signature of the informed consent, regardless of the completion of all the screening procedures.

A subject will be defined as <u>eligible</u> if he/she meets all the inclusion/exclusion criteria. Otherwise he/she will be defined as a <u>screen failure</u>.

A subject will be defined as <u>enrolled</u> in the study if he/she is included into the interventional phase of the study. The enrolment will be performed through randomised allocation to one treatments sequence.

An eligible but not enrolled subject will be defined as a reserve.

A subject will be defined as <u>randomised</u> in the study when he/she is assigned to a randomised treatments sequence.

The following analysis sets are defined:

- *Enrolled Set*: all enrolled subjects. This analysis set will be used for demographic, baseline and background characteristics
- Safety Set: all subjects who receive at least one dose of the investigational medicinal products. This analysis set will be used for the safety analyses
- *PK Set*: all randomised subjects who fulfil the study protocol requirements in terms of investigational medicinal product intake and have evaluable PK data readouts for the planned treatment comparisons, with no major deviations that may affect the PK results. This analysis set will be used for the statistical analysis of the PK results

Each subject will be coded by the CRO Biometry Unit as valid or not valid for the Safety set and the PK set. Subjects will be evaluated according to the treatment they actually receive.

# 8.2.1.1 Reasons for exclusion from the PK Set before bioanalysis

Reasons for the exclusion of subjects from the PK set are the following:

- vomiting and diarrhoea after drug intake which could render the plasma concentrationtime profile unreliable
- intake of concomitant medications which could render the plasma concentration-time profile unreliable
- AEs which could render the plasma concentration-time profile unreliable
- administration errors which could render the plasma concentration-time profile unreliable
- other events which could render the plasma concentration-time profile unreliable

If one of these events occurs, it will be noted in the CRF as the study is being conducted.



# 8.2.1.2 Reasons for exclusion from the PK Set after bioanalysis

Exclusion of subjects on the basis of pharmacokinetic reasons is possible only for:

- subjects with lack of any measurable concentrations or only very low plasma concentrations for the reference medicinal product. A subject is considered to have very low plasma concentrations if his/her AUC is less than 5% of the reference medicinal product geometric mean AUC (which should be calculated without inclusion of data from the outlying subject)
- subjects with implausible concentrations (i.e. different from the known, expected concentration profiles) for the reference medicinal product. The exclusion of these subjects must be justified on the basis of sound scientific reasons and mutually agreed between the CRO and the Sponsor
- subjects with non-zero baseline concentrations > 5% of  $C_{max}$

The samples from the subjects excluded from the PK set should still be assayed and the results listed. Subjects should not be excluded from the PK set if the  $AUC_{0-t}$  covers less than 80% of the  $AUC_{0-\infty}$ .

# 8.3 Sample size and power considerations

Data from previous PK studies of the test product, 1897 and 162020 (see the study protocol (5) for further details) were used to calculate the sample size of the present study, as shown in the table below.

**Table 9.4.1 - Sample size calculation** 

| Parameter | δ | $CV_{WR}$ | α | β | n | N=2n |
|--------------------|--------|-----------|-----|-----|----|------|
| $C_{max}$ | 1.11 | 0.3266 | 0.1 | 0.2 | 26 | 52 |
| AUC <sub>0-t</sub> | 1.0917 | 0.1265 | 0.1 | 0.2 | 4 | 9 |

 $\delta$ : ratio of geometric means of the considered parameter; CVwr%: within-subject variability;  $\alpha$ : type 1 error;  $\beta$ : type 2 error; n: number of subjects per sequence; N: total sample size

Variability of AUC<sub>0-t</sub> and C<sub>max</sub> (CVwr) actually observed in study 162020 (§ 1.4.2) was used in the calculation. The actual ratio of geometric means of AUC<sub>0-t</sub> of study 162020 was 1.0917, whilst that of C<sub>max</sub> observed in study 162020 was 1.1582. This high ratio did not prevent the demonstration of bioequivalence of the formulations in study 162020 also for C<sub>max</sub>. However, the calculation of the sample size for the present study using a  $\delta$  of 1.1582 would be 126 subjects. Considering that the enrolment of at least 126 subjects in a bioequivalence study would be hardly justifiable, that bioequivalence between the test IMP and Rilutek® 50 mg tablets available in US was demonstrated in study 162020 in 30 subjects, who completed the study, and t hat t he a ctual  $\delta$  o f C max obtained in the previous pilot study 1897 was 0.9436, which is notably nearer the equality, i.e. ratio = 1.00, than the ratio 1.1582 observed later in study 162020, a ratio of 1.11 was postulated in the present sample size calculation. Indeed, maintaining CVwr,  $\alpha$  and  $\beta$  unchanged and assuming as C<sub>max</sub> ratios, alternately, 1.05 and 1.10, sample sizes of 26 and 46 subjects, respectively, would be necessary to demonstrate bioequivalence in terms of C<sub>max</sub>.

Taking into account this premise, when the sample size in each sequence group is 26 (and the



total sample size is 52), a replicate crossover design will have 80% power to reject both the null hypothesis that the ratio of the test mean to the reference mean of  $C_{max}$  is below 0.800 and the null hypothesis that the ratio of test mean to the reference mean of  $C_{max}$  is above 1.250 (i.e. that the test and standard are not equivalent, in favour of the alternative hypothesis that the means of the two treatments are equivalent) assuming that data will be analysed in the natural log scale using t-tests for differences in means and that each t-test will be made at the 5.0% significance level.

In conclusion, 54 subjects will be enrolled in order to have 52 completed subjects.

# 8.4 Demographic, baseline and background characteristics

Demographic, baseline and background characteristics will be reported for all the enrolled subjects and analyses will be performed according to the treatment they actually received (Safety Set and PK Set).

# 8.4.1 Subjects' disposition

The disposition of all subjects enrolled in the study will be listed (Listing 16.2.4.1) and summarised (Table 14.1.1.1). The number and proportion of subjects enrolled, randomised, treated and completing the study, the number and proportion of withdrawals and the reasons for withdrawal will be presented.

# 8.4.2 Analysis sets

The subjects included in each analysis sets will be listed (Listing 16.2.4.2) and summarised (Table 14.1.1.2) by treatment group.

# 8.4.3 Subjects excluded from PK and /or safety analysis

All subjects excluded from the PK and /or safety analysis will be listed (Listing 16.2.3.1) and the reasons for exclusion will be reported.

# 8.4.4 Discontinued subjects

All subjects who discontinued the clinical trial (if any) will be listed (Listing 16.2.1.1). Last IMP administered before discontinuation, gender, age, last visit performed before discontinuation, time elapsed from last IMP administration (days), date of premature discontinuation and primary reason for subject premature discontinuation will be reported.

#### 8.4.5 Protocol deviations

All the protocol deviations reported during the clinical trial will be listed (Listing 16.2.2.1) and summarised by severity (major and minor) (Table 14.1.1.5). The number and proportion of subjects for each deviation will be reported.



# 8.4.6 Demography

Demographic data will be listed (Listing 16.2.4.3) and summarised (Table 14.1.1.3). The number and proportion of subjects in each category for categorical variables (e.g. race) and descriptive statistics (mean, SD, CV%, minimum, median and maximum) for continuous variables (e.g. age, weight) will be presented.

#### 8.4.7 Inclusion/exclusion criteria not met

All the unmet inclusion/exclusion criteria will be listed (Listing 16.2.4.4) and summarised (Table 14.1.1.4).

#### 8.4.8 ECG

The date/time of ECG assessments, the value of parameters and the overall investigator's interpretation (as normal, abnormal, not clinically significant or abnormal, clinically significant) will be listed (Listing 16.2.4.5).

The overall investigator's interpretations will be summarised using contingency tables at screening (Table 14.1.1.6).

# 8.4.9 Medical and surgical history

All the diseases of medical history and the surgeries of all subjects enrolled in the study will be coded using the Medical Dictionary for Regulatory Activities (MedDRA) version 24.0, listed (Listing 16.2.10.1).

# 8.4.10 Prior and concomitant medication

All prior and concomitant medications will be coded using the World Health Organization Drug Dictionary Enhanced (WHODDE) March 2021 and listed (Listing 16.2.10.4).

# 8.4.11 Subjects' study visits

The dates of all subjects study visits and date/time of home discharge at the end of each period will be listed (Listing 16.2.10.5).

#### 8.4.12 Fertility status and contraceptive method

The fertility status and the contraceptive method used by the subjects will be listed (Listing 16.2.10.6).

# 8.4.13 Alcohol breath test, pregnancy test, cotinine test and urine drug test

The date/time and the result of alcohol breath test, pregnancy test, cotinine test and urine drug test will be listed (Listing 16.2.8.1).



# 8.4.14 Tobacco consumption

Individual tobacco consumption habits history collected at screening will be listed (Listing 16.2.4.6).

#### **8.4.15** Meals

The start date/time of the standardised meals will be listed (Listing 16.2.10.7).

#### 8.5 IMP administration

The date and time of all IMP administrations, of film dissolution, of accidental film swallowing and reference tablet administrations will be listed (Listing 16.2.5.1). Dosing time is defined as the time the film is placed on the subject's tongue.

The actual time of film dissolution will be summarised by descriptive statistics (Table 14.2.4.1).

# 8.5.1 Dose per body weight

The dose per body weight of riluzole will be listed (Listing 16.2.5.2) and summarised using descriptive statistics (Table 14.3.5.5).

The body weight collected at the screening visit will be used for the calculation.

#### 8.5.2 Wash-out

The minimum and maximum number of days of wash-out between periods will be presented (Table 14.3.5.6).

# 8.6 PK and Palatability analysis

The date/time and score of palatability (for test only) will be listed (Listing 16.2.6.2) and summarised in tables of frequency (Table 14.2.4.2) on the safety set.

The PK analysis will be performed on the subjects included into the PK Set. Subjects will be analysed according to the treatment they actually received.

# 8.6.1 PK blood samples collection

The actual date/time of PK blood samples collection will be listed (Listing 16.2.5.3).

# 8.6.2 Descriptive pharmacokinetics/pharmacodynamics

A descriptive PK will be presented.

Individual subject concentrations of riluzole will be presented in data listings (Listing 16.2.5.4) and summarised at each time point by treatment (Table 14.2.1.1).



Individual (figures in section 16.2.5) and mean curves (+SD at sampling times) (figures in section 14.2.1), indicating inter-subject variability, will be plotted. Mean curves will be presented by treatment.

PK parameters of riluzole will be listed (Listing 16.2.6.1) and summarised by treatment (Table 14.2.2.1).

Data below the lower quantification limit (BLQL) will be considered as 0 in the calculations and presented as BLQL in listings and tables. As a consequence of BLQL (i.e. 0) values, calculated geometric means (if requested) could be null. For this reason, in the presence of any null value, the geometric mean will be reported as NC. If for an individual PK curve, a log-linear regression with a correlation coefficient  $R^2 > 0.8$  cannot be obtained, the extrapolated PK parameters will be reported as NC and considered missing in the calculations of descriptive statistics.

#### 8.6.3 Statistical comparison of pharmacokinetic parameters

According to the current European Guideline on the Investigation of Bioequivalence (3), plasma riluzole  $AUC_{0-t}$ ,  $AUC_{0-\infty}$  and  $C_{max}$  will be analysed using analysis of variance (ANOVA) (Table 14.2.3.1).

A mixed linear model will be used to make statistical inferences about the values of  $C_{\text{max}}$  and  $AUC_{0-t}$ . In order to correctly assume normality and homoscedasticity, the data will be transformed prior to analysis using a neperian logarithmic transformation in compliance with the EMA guideline.

The 90% CI of the ratio of the population means (test/reference), for the parameters under consideration will be calculated. This method is equivalent to the corresponding two one-sided test procedure with the null hypothesis of bioequivalence at the 5% significance level.

- The statistical analysis will take into account treatment, period, sequence and subject within sequence as fixed effects.
- Acceptance criterion for bioequivalence in terms of extent of absorption (AUC<sub>0-t</sub> as primary variable and AUC<sub>0-∞</sub> as secondary variable) will be that the 90% CI of this ratio has to lie within the range 80.00-125.00%.
- Due to the replicate design of the study, if the within-subject variability ( $CV_{WR}\%$ ) of  $C_{max}$  of plasma riluzole after administration of the reference formulation is >30%, the reference-scaled BE approach will be used. Bioequivalence acceptance range for  $C_{max}$  will be widened, in compliance with the guideline, as exemplified in Table 8.9.3.1.
- $CV_{WR}\%$  will be calculated by applying the formula  $CV_{WR}(\%) = 100\sqrt{e^{S^2_{WR}} 1}$ , where  $S^2_{WR}$  is the within-subject variation plasma riluzole after administration of the reference formulation only.
- The extent of the widening will be defined on the basis of the within-subject variability actually observed in the study according to  $[U, L] = \exp\left[\pm k \cdot S_{WR}\right]$ , where U is the upper limit of the acceptance range, L is the lower limit of the acceptance range, k is the regulatory constant set to 0.760 and  $S_{WR}$  is the within-subject standard deviation of the log-transformed values of  $C_{max}$  of plasma riluzole after administration of the reference formulation.



Table 8.9.3.1 Examples of widened bioequivalence acceptance limits of C<sub>max</sub> according to its actual CV<sub>WR</sub>

| CV <sub>WR</sub> %* | Lower Limit | Upper Limit |
|---------------------|-------------|-------------|
| 30 | 80.00 | 125.00 |
| 35 | 77.23 | 129.48 |
| 40 | 74.62 | 134.02 |
| 45 | 72.15 | 138.59 |
| ≥50 | 69.84 | 143.19 |

<sup>\*:</sup>  $CVWR(\%) = 100\sqrt{e^{S^2_{WR}} - 1}$ ; source: reference (3)

The value of within-subject variability of  $C_{max}$  (after administration of the reference formulation), obtained using the formula above, will be reported in the table 14.2.3.2.

 $t_{max}$  and  $t_{1/2}$  will be compared between treatments by the non-parametric Friedman test (Table 14.2.3.3).

# 8.7 Safety and tolerability analysis

The safety and tolerability analysis will be performed on the subjects included into the Safety Set.

Subjects will be analysed according to the treatment they actually received.

#### 8.7.1 Adverse events

Adverse events (AEs) will be coded by System Organ Class (SOC) and Preferred Term (PT), using the Medical Dictionary for Regulatory Activities (MedDRA).

AEs will be classified as pre-treatment AEs (PTAEs) and treatment-emergent AEs (TEAEs), according to the period of occurrence, as follows:

- PTAEs: all AEs occurring before the first dose of IMP and not worsening after the first dose of IMP
- TEAEs: all AEs occurring or worsening after the first dose of IMP

Individual PTAEs and TEAEs will be listed in subject data listings (Listing 16.2.7.1, Listing 16.2.7.2).

No summary table will be provided for PTAEs.

TEAEs will be summarised by treatment group and overall. The number and percentage of subjects with any TEAE and the number of TEAEs will be tabulated by SOC and PT, seriousness, relationship to treatment and severity.

For TEAEs that change intensity during the study (e.g. from mild to moderate or from moderate to mild), the most severe intensity will be reported in the summary tables (Table 14.3.1.1, Table 14.3.1.2, Table 14.3.1.3, Table 14.3.1.4).

Should any serious TEAE occur, the number and percentage of subjects with any serious TEAE, the number of serious TEAEs, the number and percentage of subjects with any serious



TEAE related to study drug and the number of serious TEAEs related to study drug will be presented (Table 14.3.1.5, Table 14.3.1.6).

All TEAEs leading to death will be listed, all Serious TEAEs will be listed and all TEAEs leading to discontinuation will be listed, if applicable (Table 14.3.2.1).

# 8.7.2 Vital signs

The date/time of vital signs assessments and the values of vital signs will be listed (Listing 16.2.9.1) and summarised using descriptive statistics at screening and end of study (Table 14.3.5.2) and by treatment during the study (Table 14.3.5.3).

A table of all the abnormal vital signs' values will be presented (Table 14.3.5.1).

# 8.7.3 Laboratory data

Date/time of samples collection and all laboratory results will be listed (Listing 16.2.8.1) and a table of all the abnormal values will be presented (Table 14.3.4.1).

Overall Investigator's interpretation (as normal or abnormal and, if abnormal, clinically significant or not clinically significant) and clinically significant findings (if any) will be listed (Listing 16.2.8.2).

The overall Investigator's interpretation will be summarised using tables of frequency (Table 14.3.4.2).

# 8.7.4 Physical examination

Date of the physical examination, overall Investigator's interpretation (as normal or abnormal and, if abnormal, clinically significant or not clinically significant) and clinically significant abnormalities (if any) will be listed (Listing 16.2.10.2).

# 8.7.5 Mouth Visual Inspection

The date/time of mouth visual inspection, overall Investigator's interpretation (as normal or abnormal and, if abnormal, clinically significant or not clinically significant) and clinically significant abnormalities (if any) will be listed (Listing 16.2.10.3).

The overall Investigator's interpretation will be summarised using tables of frequency (Table 14.3.5.4) at each time point.

# 8.8 Analysis datasets

Analysis datasets will be created according to the version 2.1 of the ADaM model of CDISC (13).



#### 9 REFERENCES

- 1 ICH Topic E6 (R2): Good clinical practice.
- 2 ICH Topic E9: Statistical principles for clinical trials.
- Guidance on the investigation of bioequivalence. CPMP/EWP/QWP/1401/98 Rev. 1/Corr \*\*, 20 January 2010
- 4 Questions & Answers: Positions on specific questions addressed to the pharmacokinetics working party. EMA/618604/2008 Rev. 8, 10 October 2013
- Radicioni M. Protocol CRO-PK-20-344. "Comparative bioavailability study of a new riluzole orodispersible film vs. a marketed oral reference (Rilutek<sup>®</sup> tablets) in healthy male and female volunteers". Final version 1.0, 28APR2020, CROSS Research, Switzerland, 2020
- Radicioni M. Protocol amendment CRO-PK-20-344. "Comparative bioavailability study of a new riluzole orodispersible film vs. a marketed oral reference (Rilutek® tablets) in healthy male and female volunteers". Final version 1.0, 17FEB2021, CROSS Research, Switzerland, 2020
- 7 Riluzole orodispersible film. Investigator's Brochure, Edition 3.0, Aquestive Therapeutics
- 8 Rilutek SmPC, Rilutek EPAR 14 August 2019 EMEA/H/C/000109 IAIN/0060, last updated 11 November 2019
- 9 European Public Assessment Report (EPAR), Rilutek. EMEA/H/C/109
- U.S. Department of Health and Human Services and U.S. Department of Agriculture, Nutrition and your health: 2015-2020 Dietary Guidelines, Appendix 9
- 11 SAS/STAT® User's Guide
- 12 Phoenix 1.3 User's Guide, Pharsight Corporation
- 13 CDISC Analysis Data Model Version 2.1





# 10 APPENDICES

- 1. Section 14 Tables and Figures Shells
- 2. Section 16.2 Individual Subject Data Listings and Figures Shells



#### **Section 14 - Tables Shells**

| Table 14.1.1.1 - Subjects' | disposition - Enrolled set |
|----------------------------|----------------------------|
|----------------------------|----------------------------|

- Table 14.1.1.2 Analysis sets Enrolled set
- Table 14.1.1.3 Demography Enrolled set, Safety set and PK set
- Table 14.1.1.4 Inclusion/exclusion criteria not met Enrolled set, Safety set, PK set
- Table 14.1.1.5 Protocol deviations Enrolled set, Safety set and PK set
- Table 14.1.1.6 Contingency tables of investigator's interpretation of ECG at screening Enrolled set
- Table 14.2.1.1 Riluzole concentrations (ng/mL) measured in plasma PK Set
- Table 14.2.2.1 Riluzole plasma PK parameters PK Set
- Table 14.2.3.1 Statistical analysis on Riluzole plasma PK parameters PK set
- Table 14.2.3.2 Within-subject variability of C<sub>max</sub> (after administration of the reference formulation) PK Set
- Table 14.2.3.3 Non-parametric Friedman test on  $t_{max}$  and  $t_{1/2}$  PK set
- Table 14.2.4.1 Descriptive statistics of dissolution time Safety set
- Table 14.2.4.2 Contingency tables of palatability Safety set
- Table 14.3.1.1 Global incidence of subjects with treatment-emergent adverse events Safety set
- Table 14.3.1.2 Subjects with treatment-emergent adverse events by system organ class and preferred term Safety set
- Table 14.3.1.3 Subjects with treatment-emergent adverse events by intensity, system organ class and preferred term Safety set
- Table 14.3.1.4 Subjects with treatment-emergent adverse events related to the IMP by system organ class and preferred term Safety set
- Table 14.3.1.5 Subjects with serious treatment-emergent adverse events by system organ class and preferred term Safety set
- Table 14.3.1.6 Subjects with serious treatment-emergent adverse events related to the IMP by system organ class and preferred term Safety set
- Table 14.3.2.1 Treatment emergent adverse events leading to death, serious adverse events or treatment emergent adverse events leading to discontinuation Safety set
- Table 14.3.4.1 Abnormal laboratory values Safety set
- Table 14.3.4.2 Contingency tables of investigator's interpretation of laboratory test results Safety set
- Table 14.3.5.1 Abnormal vital signs Safety set
- Table 14.3.5.2 Descriptive statistics of vital signs and body weight at screening and end of study Safety set
- Table 14.3.5.3 Descriptive statistics of vital signs during the study Safety set
- Table 14.3.5.4 Contingency tables of investigator's interpretation of mouth visual inspection during the study Safety set
- Table 14.3.5.5 Descriptive statistics of dose per body weight Safety set
- Table 14.3.5.6 Descriptive statistics of wash-out Safety set

CROSS Research S.A. Page 1



#### Table 14.1.1.1 - Subjects' disposition - Enrolled set

| | Overall<br>n (%) |
|--------------------------------------------|------------------|
| Enrolled | nn |
| Enrolled but not randomised <sup>1</sup> | nn(xx.x) |
| Randomised <sup>1</sup> | nn(xx.x) |
| Discontinued before treatment <sup>2</sup> | nn(xx.x) |
| Treated <sup>2</sup> | nn (xx.x) |
| Completed <sup>3</sup> | nn (xx.x) |
| Discontinued <sup>3</sup> | nn (xx.x) |
| Adverse event <sup>3</sup> | nn(xx.x) |
| Withdrawal by subject <sup>3</sup> | nn (xx.x) |
| | nn (xx.x) |

Note: The number and the proportion of subjects of each disposition event are reported

Note 1: The denominator for calculating the proportion is the number of enrolled subjects

Note 2: The denominator for calculating the proportion is the number of randomised subjects

Note 3: The denominator for calculating the proportion is the number of randomised and treated subjects

Source: Listing 16.2.4.1 - Subjects' disposition

Program: Tables\k344-ds-tbl.sas

CROSS Research S.A.



Table 14.1.1.2 - Analysis sets - Enrolled set

| | Riluzole 50 mg<br>orodispersible film (T)<br>N=XX<br>n (%) | Enrolled Set Rilutek®, 50 mg riluzole tablets (R) N=XX n (%) | Overall<br>N=XX<br>n (%) |
|---|---|---|---|
| Safety Set | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| PK Set | nn (xx.x) | nn (xx.x) | nn (xx.x) |

Note: Subjects are summarised according to the product they were assigned to

The number and the proportion of subjects included in each analysis set are reported

The denominator for calculating the proportions is the number of subjects in the enrolled set of each treatment group and overall

Source: Listing 16.2.4.2 - Analysis sets

Program: Tables\k344-ds-tbl.sas

CROSS Research S.A.


Table 14.1.1.3 - Demography - Enrolled set, Safety set and PK set

| | | Statistics | Enrolled Set<br>N=XX | Safety Set<br>N=XX | PK Set<br>N=XX |
|---|---|---|---|---|---|
| Sex | Female | n (%) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| | Male | n (%) | nn(xx.x) | nn (xx.x) | nn (xx.x) |
| Race | American Indian or Alaska Native | n (%) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| | Asian | n (%) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| | Native Hawaiian or Other Pacific Islander | n (%) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| | Black or African American | n (%) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| | White | n (%) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| | Other | n (%) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| Age (years) | | N | nn | nn | nn |
| | | Mean | XX.X | XX.X | XX.X |
| | | SD | XX.X | XX.X | XX.X |
| | | CV% | XX.X | XX.X | XX.X |
| | | Min | XX | XX | XX |
| | | Median | XX.X | XX.X | XX.X |
| | | Max | XX | XX | XX |
| Body Weight (kg) | | N | nn | nn | nn |
| , , , , | | Mean | XX.XX | XX.XX | XX.XX |
| | | SD | XX.XX | XX.XX | XX.XX |
| | | CV% | XX.XX | XX.XX | XX.XX |
| | | Min | XX.X | XX.X | XX.X |
| | | Median | XX.XX | XX.XX | XX.XX |
| | | Max | XX.X | XX.X | XX.X |

Note: The number and the proportion of subjects of each sex and race are reported

The denominator for calculating the proportions is the number of subjects in each analysis set

Source: Listing 16.2.4.3 - Demography

Program: Tables\k344-dm-tbl.sas



Table 14.1.1.3 - Demography - Enrolled set, Safety set and PK set

| | Statistics | Enrolled Set<br>N=XX | Safety Set<br>N=XX | PK Set<br>N=XX |
|---|---|---|---|---|
| Body Mass Index (kg/m²) | N | nn | nn | nn |
| | Mean | XX.XX | XX.XX | XX.XX |
| | SD | XX.XX | XX.XX | XX.XX |
| | CV% | XX.XX | XX.XX | XX.XX |
| | Min | XX.X | XX.X | XX.X |
| | Median | XX.XX | XX.XX | XX.XX |
| | Max | XX.X | XX.X | XX.X |

Note: The number and the proportion of subjects of each sex and race are reported

The denominator for calculating the proportions is the number of subjects in each analysis set

Source: Listing 16.2.4.3 - Demography Program: Tables\k344-dm-tbl.sas



Table 14.1.1.4 - Inclusion/exclusion criteria not met - Enrolled set, Safety set, PK set

| | Enrolled Set<br>N=XX | Safety Set<br>N=XX | PK Set<br>N=XX |
|---|---|---|---|
| Number of subjects with any inclusion/exclusion criteria not met | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| Inclusion | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| Inclusion criterion 1 Inclusion criterion 2 | | nn (xx.x)<br>nn (xx.x) | nn (xx.x)<br>nn (xx.x) |
| Exclusion | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| Exclusion criterion 1 Exclusion criterion 2 | nn (xx.x)<br>nn (xx.x) | nn (xx.x)<br>nn (xx.x) | nn (xx.x)<br>nn (xx.x) |

Note: The number and the proportion of subjects for any criterion not met are reported

The denominator for calculating the proportions is the number of subjects in each analysis set

Source: Listing 16.2.4.4 - Inclusion/Exclusion criteria not met

 $Program: Tables \verb|\k344-ie-tbl.sas|$ 



Table 14.1.1.5 - Protocol deviations - Enrolled set, Safety set, PK set

| | Enrolled Set<br>N=XX | Safety Set<br>N=XX | PK Set<br>N=XX |
|---|---|---|---|
| Number of subjects with any protocol deviation | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| Major | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| Treatment deviation | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| Inclusion criteria violation | nn(xx.x) | nn(xx.x) | nn (xx.x) |
| Exclusion criteria violation | nn(xx.x) | nn(xx.x) | nn(xx.x) |
| Medication not admitted | nn(xx.x) | nn(xx.x) | nn(xx.x) |
| Minor | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| Deviation from scheduled sampling time | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| | | ••• | |

Note: The number and the proportion of subjects for any protocol violation are reported

The denominator for calculating the proportions is the number of subjects in each analysis set

Source: Listing 16.2.2.1 - Protocol deviations

Program: Tables\k344-dv-tbl.sas



Table 14.1.1.6 - Contingency tables of investigator's interpretation of ECG at screening - Enrolled set

| Time Point | Investigator's interpretation | Enrolled Set<br>N=XX |
|------------|--------------------------------------|----------------------|
| Screening | Normal | nn (xx.x) |
| | Abnormal, Not Clinically Significant | nn(xx.x) |
| | Abnormal, Clinically Significant | nn (xx.x) |

Note: The number and the proportion of subjects for each classification level are reported

The denominator for calculating the proportions is the number of subjects in the enrolled set

Source: Listing 16.2.4.5 - Investigator's interpretation of ECG

Program: Tables\k344-eg-tbl.sas



Table 14.2.1.1 - Riluzole concentrations (ng/mL) measured in plasma - PK Set

Investigational Medicinal Product: Riluzole 50 mg orodispersible film (T)

| Statistics | Pre<br>dose | 0.25 h | 0.5 h | 0.75 h | 1 h | 1.25 h | 1.5 h | 2 h | 3 h | 4 h | 6 h | 8 h | 12 h | 18 h | 24 h |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| N | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| Geo.Mean | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX |
| Mean | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX |
| SD | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX |
| CV% | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX |
| Min | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X |
| Median | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX |
| Max | xxx.x | xxx.x | XXX.X | xxx.x | xxx.x | xxx.x | XXX.X | XXX.X | xxx.x | xxx.x | xxx.x | xxx.x | xxx.x | xxx.x | XXX.X |

BLQL: Below Lower Quantification Limit (x.xx ng/mL)

Source: Listing 16.2.5.4 - Riluzole concentrations (ng/mL) measured in plasma

Program: pk-analysis\k344-tlf.sas



Table 14.2.1.1 - Riluzole concentrations (ng/mL) measured in plasma - PK Set

Investigational Medicinal Product: Rilutek®, 50 mg riluzole tablets (R)

| Statistics | Pre<br>dose | 0.25 h | 0.5 h | 0.75 h | 1 h | 1.25 h | 1.5 h | 2 h | 3 h | 4 h | 6 h | 8 h | 12 h | 18 h | 24 h |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| N | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| Geo.Mean | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX |
| Mean | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX |
| SD | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX |
| CV% | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX |
| Min | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X |
| Median | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX |
| Max | xxx.x | XXX.X | XXX.X | xxx.x | xxx.x | xxx.x | xxx.x | XXX.X | xxx.x | xxx.x | xxx.x | xxx.x | xxx.x | xxx.x | XXX.X |

BLQL: Below Lower Quantification Limit (x.xx ng/mL)

Source: Listing 16.2.5.4 - Riluzole concentrations (ng/mL) measured in plasma

 $Program: pk-analysis \backslash k344-tlf.sas$ 



Table 14.2.2.1 - Riluzole plasma PK parameters - PK Set

Investigational Medicinal Product: Riluzole 50 mg orodispersible film (T)

| Statistics | C <sub>max</sub><br>(ng/mL) | t <sub>max</sub><br>(h) | AUC <sub>0-t</sub> (h*ng/mL) | $\begin{array}{c} AUC_{0\text{-}inf} \\ (h*ng/mL) \end{array}$ | t½<br>(h) | $\lambda_z$ (1/h) |
|---|---|---|---|---|---|---|
| N | XX | XX | XX | XX | XX | XX |
| Geo.Mean | XXX.XX | xxx.xx | xxx.xx | XXX.XX | xxx.xx | XXX.XX |
| Mean | XXX.XX | xxx.xx | xxx.xx | XXX.XX | xxx.xx | XXX.XX |
| SD | XXX.XX | xxx.xx | xxx.xx | XXX.XX | xxx.xx | XXX.XX |
| CV% | XXX.XX | XXX.XX | xxx.xx | XXX.XX | xxx.xx | XXX.XX |
| Min | XXX.XX | xxx.xx | XXX.XX | XXX.XX | xxx.xx | XXX.XX |
| Median | XXX.XX | XXX.XX | xxx.xx | XXX.XX | xxx.xx | XXX.XX |
| Max | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX | XXX.XX |

Source: Listing 16.2.6.1 - Riluzole plasma PK parameters

 $Program: pk-analysis \backslash k344-tlf.sas$ 



Table 14.2.2.1 - Riluzole plasma PK parameters - PK Set

Investigational Medicinal Product: Rilutek®, 50 mg riluzole tablets (R)

| Statistics | C <sub>max</sub><br>(ng/mL) | t <sub>max</sub><br>(h) | AUC <sub>0-t</sub><br>(h*ng/mL) | AUC <sub>0-inf</sub> (h*ng/mL) | t½<br>(h) | $\lambda_z$ (1/h) |
|---|---|---|---|---|---|---|
| N | XX | XX | XX | XX | XX | XX |
| Geo.Mean | XXX.XX | XXX.XX | XXX.XX | xxx.xx | xxx.xx | XXX.XX |
| Mean | XXX.XX | XXX.XX | XXX.XX | xxx.xx | xxx.xx | XXX.XX |
| SD | XXX.XX | XXX.XX | XXX.XX | xxx.xx | xxx.xx | XXX.XX |
| CV% | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX |
| Min | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX |
| Median | XXX.XX | XXX.XX | XXX.XX | xxx.xx | xxx.xx | XXX.XX |
| Max | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX | xxx.xx |

Source: Listing 16.2.6.1 - Riluzole plasma PK parameters

 $Program: pk-analysis \backslash k344-tlf.sas$ 



Table 14.2.3.1 - Statistical analysis on riluzole plasma PK parameters - PK set

| Analysis | Dependent Variable | Comparison | Point Estimate | 90% Confidence Interval<br>Lower Limit | 90% Confidence Interval<br>Upper Limit | Effect | p Value |
|---|---|---|---|---|---|---|---|
| ANOVA | Ln(AUC <sub>0-inf</sub> ) | T vs R | xxx.xx | xxx.xx | xxx.xx | Sequence<br>Treatment<br>Period | x.xxxx<br>x.xxxx<br>x.xxxx |
| ANOVA | Ln(AUC <sub>0-t</sub> ) | T vs R | xxx.xx | xxx.xx | xxx.xx | Sequence<br>Treatment<br>Period | XXXXX<br>X.XXXX<br>X.XXXX |
| ANOVA | Ln(C <sub>max</sub> ) | T vs R | xxx.xx | xxx.xx | XXX.XX | Sequence<br>Treatment<br>Period | x.xxxx<br>x.xxxx<br>x.xxxx |

T: Riluzole 50 mg orodispersible film (T)

R: Rilutek®, 50 mg riluzole tablets (R) \_

 $Program: pk-analysis \backslash k344-tlf.sas$ 





Table 14.2.3.2 - Within-subject variability of  $C_{max}$  (after administration of the reference formulation) - PK Set

| AINGR | Dependent Variable | ${ m S^2_{WR}}$ | Within-subject variability |
|----------|--------------------|-----------------|----------------------------|
| | | | CV <sub>WR</sub> (%) |
| Riluzole | $Ln(C_{max})$ | xxx.xxx | XX.XX |

Note:  $CV_{WR}\%$  was calculated by applying the formula  $100*sqrt[exp(S^2_{WR})-1]$ 

 $Program: pk-analysis \backslash k344-tlf.sas$ 



Table 14.2.3.3 - Non-parametric Friedman test on  $t_{max}$  and  $t_{1/2}$  - PK set

| Analysis | Dependent Variable | Comparison | p Value |
|----------|---------------------------|------------------|------------------|
| Friedman | $t_{ m max}$ $t_{ m 1/2}$ | T vs R<br>T vs R | X.XXXX<br>X.XXXX |

Program: pk-analysis\k344-tlf.sas



Table 14.2.4.1 - Descriptive statistics of dissolution time (Safety set)

| | | | Safety Set | |
|---|---|---|---|---|
| | | Statistics | Riluzole 50 mg<br>orodispersible film (T)<br>1 <sup>st</sup> adm.<br>N=XX | Riluzole 50 mg<br>orodispersible film (T)<br>2 <sup>nd</sup> adm.<br>N=XX |
| Was the film accidentally swallowed within 5 min after dosing? | Yes | n (%) | nn (xx.x) | nn (xx.x) |
| | No | n (%) | nn (xx.x) | nn (xx.x) |
| Was the film undissolved at 5 min after dosing and had to be swallowed? | Yes | n (%) | nn (xx.x) | nn (xx.x) |
| | No | n (%) | nn (xx.x) | nn (xx.x) |
| Dissolution Time [min] | | N | nn | nn |
| | | Mean | XXX.XX | XXX.XX |
| | | SD | XXX.XX | XXX.XX |
| | | CV% | XXX.XX | XXX.XX |
| | | Min | XXX.X | XXX.X |
| | | Median | XXX.XX | XXX.XX |
| | | Max | XXX.X | XXX.X |

Note: Subjects are summarised according to the product they actually received

The number and the proportion of subjects for each question are reported

The denominator for calculating the proportions is the number of subjects in the safety set of Riluzole 50 mg orodispersible film (T) of each administration

Source: Listing 16.2.5.1 - Investigational medicinal products administration

 $Program: Tables \backslash k344\text{-}ex\text{-}tbl.sas$ 



Table 14.2.4.2 - Contingency tables of palatability - Safety set

| | | Safet | Safety Set |
|---|---|---|---|
| Time Point | Palatability Score | Riluzole 50 mg<br>orodispersible film (T)<br>1 <sup>st</sup> adm.<br>N=XX | Riluzole 50 mg<br>orodispersible film (T)<br>2 <sup>nd</sup> adm.<br>N=XX |
| Immediately after administration | 0 - very unpleasant | xx (xx.x) | nn (xx.x) |
| | 1 - unpleasant | xx (xx.x) | nn (xx.x) |
| | 2 - acceptable | xx (xx.x) | nn (xx.x) |
| | 3 - good | xx (xx.x) | nn (xx.x) |
| | 4 - very good | xx (xx.x) | nn (xx.x) |

Note: The number and the proportion of subjects for each classification level are reported

The denominator for calculating the proportions is the number of subjects in the safety set of Riluzole 50 mg orodispersible film (T) of each administration

Source: Listing 16.2.6.2 - Palatability Program: Tables\k344-fa-tbl.sas



Table 14.3.1.1 - Global incidence of subjects with treatment-emergent adverse events - Safety set

| | Riluzole 50 mg<br>orodispersible film (T)<br>N=XX<br>n (%) [n AE] | Safety Set Rilutek®, 50 mg riluzole tablets (R) N=XX n (%) [n AE] | Overall<br>N=XX<br>n (%) [n AE] |
|---|---|---|---|
| Treatment-emergent Adverse Events | nn(xx.x)[kk] | nn (xx.x) [kk] | nn (xx.x) [kk] |
| Relationship | nn(xx.x)[kk] | nn (xx.x) [kk] | nn(xx.x)[kk] |
| Related | nn(xx.x)[kk] | nn(xx.x)[kk] | nn(xx.x)[kk] |
| Not related | nn(xx.x)[kk] | nn(xx.x)[kk] | nn(xx.x)[kk] |
| Intensity | nn(xx.x)[kk] | nn (xx.x) [kk] | nn (xx.x) [kk] |
| Mild | nn(xx.x)[kk] | nn(xx.x)[kk] | nn (xx.x) [kk] |
| Moderate | nn(xx.x)[kk] | nn(xx.x)[kk] | nn(xx.x)[kk] |
| Severe | nn(xx.x)[kk] | nn(xx.x)[kk] | nn(xx.x)[kk] |
| Leading to discontinuation | nn(xx.x)[kk] | nn(xx.x)[kk] | nn (xx.x) [kk] |

Note: Subjects are summarised according to the product they actually received

Subjects are summarised according to the each level of relationship and intensity reported in each treatment group and overall

The number and the proportion of subjects with any adverse event and the number of adverse events for each classification level are reported

The denominator for calculating the proportions is the number of subjects in the safety set of each treatment group and overall

Source: Listing 16.2.7.1 - Treatment-emergent adverse events

Program: Tables\k344-ae-01-tbl.sas



Table 14.3.1.1 - Global incidence of subjects with treatment-emergent adverse events - Safety set

| | Riluzole 50 mg<br>orodispersible film (T)<br>N=XX<br>n (%) [n AE] | Safety Set Rilutek®, 50 mg riluzole tablets (R) N=XX n (%) [n AE] | Overall<br>N=XX<br>n (%) [n AE] |
|---|---|---|---|
| Serious Treatment-emergent Adverse Events | nn (xx.x) [kk] | nn (xx.x) [kk] | nn (xx.x) [kk] |
| Relationship | nn (xx.x) [kk] | nn (xx.x) [kk] | nn (xx.x) [kk] |
| Related | nn (xx.x) [kk] | nn(xx.x)[kk] | nn (xx.x) [kk] |
| Not related | nn(xx.x)[kk] | nn(xx.x)[kk] | nn(xx.x)[kk] |
| Intensity | nn (xx.x) [kk] | nn (xx.x) [kk] | nn (xx.x) [kk] |
| Mild | nn (xx.x) [kk] | nn(xx.x)[kk] | nn(xx.x)[kk] |
| Moderate | nn (xx.x) [kk] | nn(xx.x)[kk] | nn(xx.x)[kk] |
| Severe | nn (xx.x) [kk] | nn(xx.x)[kk] | nn(xx.x)[kk] |
| Leading to discontinuation | nn (xx.x) [kk] | nn(xx.x)[kk] | nn (xx.x) [kk] |

Note: Subjects are summarised according to the product they actually received

Subjects are summarised according to the each level of relationship and intensity reported in each treatment group and overall

The number and the proportion of subjects with any adverse event and the number of adverse events for each classification level are reported

The denominator for calculating the proportions is the number of subjects in the safety set of each treatment group and overall

Source: Listing 16.2.7.1 - Treatment-emergent adverse events

 $Program: Tables \verb|\k344-ae-01-tbl.sas|$ 



Table 14.3.1.2 - Subjects with treatment-emergent adverse events by system organ class and preferred term - Safety set

| System Organ Class <sup>1</sup> Preferred Term <sup>1</sup> | Riluzole 50 mg<br>orodispersible film (T)<br>N=XX<br>n (%) [n AE] | Safety Set Rilutek®, 50 mg riluzole tablets (R) N=XX n (%) [n AE] | Overall<br>N=XX<br>n (%) [n AE] |
|---|---|---|---|
| Treatment-emergent Adverse Events | nn (xx.x) [kk] | nn (xx.x) [kk] | nn (xx.x) [kk] |
| Nervous system disorders | nn(xx.x)[kk] | nn(xx.x)[kk] | nn (xx.x) [kk] |
| Headache | nn (xx.x) [kk]<br> | nn (xx.x) [kk] | nn (xx.x) [kk] |
| Gastrointestinal disorders | nn(xx.x)[kk] | nn (xx.x) [kk] | nn(xx.x)[kk] |
| Abdominal pain upper Diarrhoea | nn (xx.x) [kk]<br>nn (xx.x) [kk]<br> | nn (xx.x) [kk]<br>nn (xx.x) [kk]<br> | nn (xx.x) [kk]<br>nn (xx.x) [kk]<br> |

Note: Subjects are summarised according to the product they actually received

The number and the proportion of subjects with any adverse event and the number of adverse events for each classification level are reported

The denominator for calculating the proportions is the number of subjects in the safety set of each treatment group and overall

Note 1: MedDRA version 24.0

Source: Listing 16.2.7.1 - Treatment-emergent adverse events

Program: Tables\k344-ae-02-tbl.sas



Table 14.3.1.3 - Subjects with treatment-emergent adverse events by intensity, system organ class and preferred term - Safety set

| | Safety Set | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| | Riluzole 50 | mg orodispers | ible film (T) | Rilutek®, | 50 mg riluzole | tablets (R) | Overall | | |
| System Organ Class <sup>1</sup> | Mild | N=XX<br>Moderate | Severe | Mild | N=XX<br>Moderate | Severe | Mild | N=XX<br>Moderate | Severe |
| Preferred Term <sup>1</sup> | n (%) [n AE] | n (%) [n AE] | n (%) [n AE] | n (%) [n AE] | n (%) [n AE] | n (%) [n AE] | n (%) [n AE] | n (%) [n AE] | n (%) [n AE] |
| Treatment-emergent Adverse Events | nn (x.x) [kk] | nn(x.x)[kk] | nn(x.x)[kk] | nn(x.x)[kk] | nn(x.x)[kk] | nn(x.x)[kk] | nn(x.x)[kk] | nn(x.x)[kk] | nn(x.x)[kk] |
| Nervous system disorders | nn(x.x)[kk] | nn(x.x)[kk] | $nn\left( x.x\right) \left[ kk\right]$ | $nn\left( x.x\right) \left[ kk\right]$ | nn(x.x)[kk] | nn(x.x)[kk] | nn(x.x)[kk] | nn(x.x)[kk] | nn(x.x)[kk] |
| Headache | nn(x.x)[kk] | nn (x.x) [kk] | nn(x.x)[kk] | nn(x.x)[kk] | nn(x.x)[kk] | nn(x.x)[kk] | nn (x.x) [kk] | nn (x.x) [kk] | nn(x.x)[kk] |
| | nn(x.x)[kk] | $nn\left( x.x\right) \left[ kk\right]$ | $nn\left( x.x\right) \left[ kk\right]$ | $nn\left( x.x\right) \left[ kk\right]$ | $nn\left( x.x\right) \left[ kk\right]$ | $nn\left( x.x\right) \left[ kk\right]$ | nn(x.x)[kk] | $nn\left( x.x\right) \left[ kk\right]$ | nn(x.x)[kk] |
| Gastrointestinal disorders | nn (x.x) [kk] | nn(x.x)[kk] | nn(x.x)[kk] | nn(x.x)[kk] | nn(x.x)[kk] | nn(x.x)[kk] | nn(x.x)[kk] | nn(x.x)[kk] | nn(x.x)[kk] |
| Abdominal pain upper | nn(x.x)[kk] | nn(x.x)[kk] | nn(x.x)[kk] | nn(x.x)[kk] | nn(x.x)[kk] | nn(x.x)[kk] | nn(x.x)[kk] | nn(x.x)[kk] | nn(x.x)[kk] |
| Diarrhoea | nn(x.x)[kk] | nn(x.x)[kk] | nn(x.x)[kk] | nn(x.x)[kk] | nn(x.x)[kk] | nn(x.x)[kk] | nn(x.x)[kk] | nn(x.x)[kk] | nn(x.x)[kk] |
| | nn(x.x)[kk] | nn(x.x)[kk] | nn(x.x)[kk] | nn(x.x)[kk] | nn(x.x)[kk] | nn(x.x)[kk] | nn(x.x)[kk] | nn(x.x)[kk] | nn(x.x)[kk] |

Note: Subjects are summarised according to the treatment they actually received

The number and the proportion of subjects with any adverse event and the number of adverse events for each classification level are reported

The denominator for calculating the proportions is the number of subjects in the safety set of each treatment group and overall

Note 1: MedDRA version 24.0

Source: Listing 16.2.7.1 - Treatment-emergent adverse events

Program: Tables\k344-ae-02-tbl.sas



Table 14.3.1.4 - Subjects with treatment-emergent adverse events related to the IMP by system organ class and preferred term - Safety set

| | | Safety Set | |
|---|---|---|---|
| System Organ Class <sup>1</sup> Preferred Term <sup>1</sup> | Riluzole 50 mg<br>orodispersible film (T)<br>N=XX<br>n (%) [n AE] | Rilutek®, 50 mg<br>riluzole tablets (R)<br>N=XX<br>n (%) [n AE] | Overall<br>N=XX<br>n (%) [n AE] |
| Treatment-emergent Adverse Events related to the IMP | nn(xx.x)[kk] | nn (xx.x) [kk] | nn (xx.x) [kk] |
| Nervous system disorders | nn(xx.x)[kk] | nn(xx.x)[kk] | nn(xx.x)[kk] |
| Headache | nn(xx.x)[kk] | nn(xx.x)[kk] | nn (xx.x) [kk] |
| | <b></b> | ••• | ••• |
| Gastrointestinal disorders | nn(xx.x)[kk] | nn(xx.x)[kk] | nn(xx.x)[kk] |
| Abdominal pain upper | nn(xx.x)[kk] | nn(xx.x)[kk] | nn(xx.x)[kk] |
| Diarrhoea | nn(xx.x)[kk] | nn(xx.x)[kk] | nn(xx.x)[kk] |
| | <b></b> | | |

Note: Subjects are summarised according to the product they actually received

The number and the proportion of subjects with any related adverse event and the number of related adverse events for each classification level are reported

The denominator for calculating the proportions is the number of subjects in the safety set of each treatment group and overall

Note 1: MedDRA version 24.0

Source: Listing 16.2.7.1 - Treatment-emergent adverse events

Program: Tables\k344-ae-02-tbl.sas



Table 14.3.1.5 - Subjects with serious treatment-emergent adverse events by system organ class and preferred term - Safety set

| | | Safety Set | |
|---|---|---|---|
| System Organ Class <sup>1</sup> Preferred Term <sup>1</sup> | Riluzole 50 mg<br>orodispersible film (T)<br>N=XX<br>n (%) [n AE] | Rilutek®, 50 mg<br>riluzole tablets (R)<br>N=XX<br>n (%) [n AE] | Overall<br>N=XX<br>n (%) [n AE] |
| Serious Treatment-emergent Adverse Events | nn(xx.x)[kk] | nn(xx.x)[kk] | nn (xx.x) [kk] |
| Nervous system disorders | nn(xx.x)[kk] | nn(xx.x)[kk] | nn(xx.x)[kk] |
| Headache | nn(xx.x)[kk] | nn(xx.x)[kk] | nn (xx.x) [kk] |
| ··· | <b></b> | <b></b> | ••• |
| Gastrointestinal disorders | nn(xx.x)[kk] | nn(xx.x)[kk] | nn(xx.x)[kk] |
| Abdominal pain upper | nn(xx.x)[kk] | nn (xx.x) [kk] | nn(xx.x)[kk] |
| Diarrhoea | nn(xx.x)[kk] | nn(xx.x)[kk] | nn(xx.x)[kk] |
| | <b></b> | | |

Note: Subjects are summarised according to the product they actually received

The number and the proportion of subjects with any serious adverse event and the number of serious adverse events for each classification level are reported

The denominator for calculating the proportions is the number of subjects in the safety set of each treatment group and overall

Note 1: MedDRA version 24.0

Source: Listing 16.2.7.1 - Treatment-emergent adverse events

Program: Tables\k344-ae-02-tbl.sas



Table 14.3.1.6 - Subjects with serious treatment-emergent adverse events related to the IMP by system organ class and preferred term - Safety set

| | Safety Set | | |
|---|---|---|---|
| System Organ Class <sup>1</sup> Preferred Term <sup>1</sup> | Riluzole 50 mg<br>orodispersible film (T)<br>N=XX<br>n (%) [n AE] | Rilutek®, 50 mg<br>riluzole tablets (R)<br>N=XX<br>n (%) [n AE] | Overall<br>N=XX<br>n (%) [n AE] |
| Serious Treatment-emergent Adverse Events related to the IMP | nn(xx.x)[kk] | nn (xx.x) [kk] | nn (xx.x) [kk] |
| Nervous system disorders | nn(xx.x)[kk] | nn(xx.x)[kk] | nn(xx.x)[kk] |
| Headache | nn (xx.x) [kk]<br> | nn (xx.x) [kk]<br> | nn (xx.x) [kk] |
| Gastrointestinal disorders | nn (xx.x) [kk] | nn (xx.x) [kk] | nn(xx.x)[kk] |
| Abdominal pain upper<br>Diarrhoea | nn (xx.x) [kk]<br>nn (xx.x) [kk] | nn (xx.x) [kk]<br>nn (xx.x) [kk] | nn (xx.x) [kk]<br>nn (xx.x) [kk] |

Note: Subjects are summarised according to the product they actually received

The number and the proportion of subjects with any serious related adverse event and the number of serious related adverse events for each classification level are reported. The denominator for calculating the proportions is the number of subjects in the safety set of each treatment group and overall

Note 1: MedDRA version 24.0

Source: Listing 16.2.7.1 - Treatment-emergent adverse events

Program: Tables\k344-ae-02-tbl.sas



Table 14.3.2.1 - Treatment emergent adverse events leading to death, serious adverse events or treatment emergent adverse events leading to discontinuation - Safety set

**Investigational Medicinal Product: Riluzole 50 mg orodispersible film (T)** 

| Subject<br>ID | Adverse<br>Event<br>ID | | |
|---|---|---|---|
| S001/001 | 1 | Description: | Headache |
| | | Body Area Affected: | Head |
| | | Preferred Term <sup>1</sup> : | Headache |
| | | System Organ Class <sup>1</sup> : | Nervous system disorders |
| | | Acknowledgment Date/Time (Day) | ddMMMyyyy hh:mm (j) |
| | | Start - End Date/Time (Day): | ddMMMyyyy hh:mm (k) - ddMMMyyyy hh:mm (k+n) |
| | | Has the Adverse Event Started After the Administration of the Study Drug? | Y |
| | | Last Study Drug Administration Date/Time Before Onset | ddMMMyyyy hh:mm |
| | | Reasonable Possibility of a Causal Relationship with the Study Drug? | Y |
| | | Other Causal Relationship | |
| | | Severity: | Severe |
| | | Pattern: | Continuous |
| | | Serious? | N |
| | | Seriousness criteria: | |
| | | Action taken with Study Drug: | None |
| | | Concomitant therapy? | N |
| | | Caused Study Discontinuation? | Y |
| | | Other Action Taken: | None |
| | | Outcome: | Recovered/Resolved |
| | | Comments: | |

Note: Subjects are listed according to the product they actually received

Note 1: MedDRA version 24.0.

Sources: Listing 16.2.7.1 - Treatment-emergent adverse events, Listing 16.2.7.2 - Pre-treatment adverse events (for serious adverse events only)

 $Program: Tables \verb+\k344-ae-03-tbl.sas$ 



Table 14.3.2.1 - Treatment emergent adverse events leading to death, serious adverse events or treatment emergent adverse events leading to discontinuation - Safety set

Investigational Medicinal Product: Rilutek®, 50 mg riluzole tablets (R)

| Subject<br>ID | Adverse<br>Event<br>ID | | |
|---|---|---|---|
| S001/001 | 2 | Description: | Headache |
| | | Body Area Affected: | Head |
| | | Preferred Term <sup>1</sup> : | Headache |
| | | System Organ Class <sup>1</sup> : | Nervous system disorders |
| | | Acknowledgment Date/Time (Day) | ddMMMyyyy hh:mm (j) |
| | | Start - End Date/Time (Day): | ddMMMyyyy hh:mm (k) - ddMMMyyyy hh:mm (k+n) |
| | | Has the Adverse Event Started After the Administration of the Study Drug? | Y |
| | | Last Study Drug Administration Date/Time Before Onset | ddMMMyyyy hh:mm |
| | | Reasonable Possibility of a Causal Relationship with the Study Drug? | Y |
| | | Other Causal Relationship | |
| | | Severity: | Severe |
| | | Pattern: | Continuous |
| | | Serious? | N |
| | | Seriousness criteria: | |
| | | Action taken with Study Drug: | None |
| | | Concomitant therapy? | N |
| | | Caused Study Discontinuation? | Y |
| | | Other Action Taken: | None |
| | | Outcome: | Recovered/Resolved |
| | | Comments: | |

Note: Subjects are listed according to the product they actually received

Note 1: MedDRA version 24.0.

Sources: Listing 16.2.7.1 - Treatment-emergent adverse events, Listing 16.2.7.2 - Pre-treatment adverse events (for serious adverse events only)

 $Program: Tables \verb|\k| 344-ae-03-tbl.sas$ 



Table 14.3.4.1 - Abnormal laboratory values - Safety set

**Category of Laboratory Parameters: BLOOD CHEMISTRY** 

| Subject<br>ID | Time<br>Point | Collection Date/time | Parameter | Value and Abnormality <sup>1</sup> | Normal Range or<br>Reference Value | Clinically<br>Significant? |
|---|---|---|---|---|---|---|
| S001/001 | Screening | ddMMMyyyy hh:mm | Phosphate [mmol/L] | 0.84 [L] | 0.87 - 1.45 | N |
| | ••• | ••• | | ••• | ••• | ••• |
| S001/001 | End of Study | ddMMMyyyy hh:mm | Phosphate [mmol/L] | 0.84 [L] | 0.87 - 1.45 | N |
| | | ••• | ··· | ••• | ••• | ••• |

Note 1: H=Higher than upper normal limit, L=Lower than lower normal limit

Source: Listing 16.2.8.1 - Individual laboratory measurements

Program: Tables\k344-lb-tbl.sas



Table 14.3.4.1 - Abnormal laboratory values - Safety set

**Category of Laboratory Parameters: HEMATOLOGY** 

| Subject<br>ID | Time<br>Point | Collection Date/time | Parameter | Value and<br>Abnormality <sup>1</sup> | Normal Range or<br>Reference Value | Clinically Significant? |
|---|---|---|---|---|---|---|
| S001/001 | Screening | ddMMMyyyy hh:mm | Leukocytes [10^9/L] | 10.02 [H] | 4.00 - 10.00 | N |
| ••• | ••• | ··· | <b></b> | | ••• | ••• |
| ••• | ••• | ••• | ••• | ••• | ••• | |
| S001/001 | End of Study | ddMMMyyyy hh:mm | Leukocytes [10^9/L] | 10.02 [H] | 4.00 - 10.00 | N |
| ••• | | | <b></b> | ••• | ••• | ••• |

Note 1: H=Higher than upper normal limit, L=Lower than lower normal limit

Source: Listing 16.2.8.1 - Individual laboratory measurements

Program: Tables\k344-lb-tbl.sas



Table 14.3.4.1 - Abnormal laboratory values - Safety set

**Category of Laboratory Parameters: URINE ANALYSIS** 

| Subject<br>ID | Time<br>Point | Collection Date/time | Parameter | Value and Abnormality <sup>1</sup> | Normal Range or Reference Value | Clinically<br>Significant? |
|---|---|---|---|---|---|---|
| S001/001 | Screening | ddMMMyyyy hh:mm | Urinary Hemoglobin | +++ [A] | Absent | N |
| <br>S001/001 | <br>End of Study | <br>ddMMMyyyy hh:mm | <br>Urinary Hemoglobin | <br>+++ [A] | <br>Absent | <br>N |
| | | ••• | <b></b> | ••• | ••• | ••• |

Note 1: A=Different from reference value

Source: Listing 16.2.8.1 - Individual laboratory measurements

Program: Tables\k344-lb-tbl.sas



Table 14.3.4.2 - Contingency tables of investigator's interpretation of laboratory test results - Safety set

| Time Point | Investigator's interpretation | Safety Set<br>N=XX |
|---|---|---|
| Screening | Normal Abnormal, Not Clinically Significant Abnormal, Clinically Significant | nn (xx.x)<br>nn (xx.x)<br>nn (xx.x) |
| End of Study | Normal Abnormal, Not Clinically Significant Abnormal, Clinically Significant | nn (xx.x)<br>nn (xx.x)<br>nn (xx.x) |

Note: The number and the proportion of subjects for each classification level are reported

The denominator for calculating the proportions is the number of subjects in the safety set

Source: Listing 16.2.8.2 - Investigator's interpretation of laboratory test results

Program: Tables\k344-lb-tbl.sas



Table 14.3.5.1 - Abnormal vital signs - Safety set

| Subject<br>ID | Time<br>Point | Assessment Date/Time | Parameter | Value and<br>Abnormality <sup>1</sup> | Normal Range | Clinically Significant? |
|---|---|---|---|---|---|---|
| S001/001 | Screening | ddMMMyyyy hh:mm | Systolic Blood Pressure [mmHg] | 96 [L] | 100-139 | N |
| S001/001 | Visit 3 - Pre-dose | ddMMMyyyy hh:mm | Systolic Blood Pressure [mmHg] | 96 [L] | 100-139 | N |
| | | | | | | ••• |

Note 1: H=Higher than upper normal limit, L=Lower than lower normal limit

Source: Listing 16.2.9.1 - Vital signs and body weight

Program: Tables\k344-vs-tbl.sas



Table 14.3.5.2 - Descriptive statistics of vital signs at screening and end of study - Safety set

| Parameter | Time Point | Statistics | Safety Set<br>N=XX |
|---|---|---|---|
| Systolic Blood Pressure [mmHg] | Screening | N | nn |
| Systolic Blood i ressure [mining] | Sciedning | Mean | |
| | | SD | XXX.X |
| | | CV% | XXX.X |
| | | | XXX.X |
| | | Min | XXX |
| | | Median | XXX.X |
| | | Max | XXX |
| Creatalia Dia ad Draggura [manalla] | End of Study | N | |
| Systolic Blood Pressure [mmHg] | End of Study | | nn |
| | | Mean | XXX.X |
| | | SD | XXX.X |
| | | CV% | XXX.X |
| | | Min | XXX |
| | | Median | XXX.X |
| | | Max | XXX |
| District Plant Day on the French Lab | G | M | |
| Diastolic Blood Pressure [mmHg] | Screening | N | nn |
| | | Mean | XXX.X |
| | | SD | XXX.X |
| | | CV% | XXX.X |
| | | Min | XXX |
| | | Median | XXX.X |
| | | Max | XXX |

Note: End of Study = Visit 9 - Day 2 - 36 hours post-dose or early termination visit for vital signs, final visit or early termination visit for body weight

Source: Listing 16.2.9.1 - Vital signs Program: Tables\k344-vs-tbl.sas



Table 14.3.5.2 - Descriptive statistics of vital signs at screening and end of study - Safety set

| Parameter | Time Point | Statistics | Safety Set<br>N=XX |
|---|---|---|---|
| Diastolic Blood Pressure [mmHg] | End of Study | N | nn |
| | | Mean | XXX.X |
| | | SD | XXX.X |
| | | CV% | XXX.X |
| | | Min | XXX |
| | | Median | XXX.X |
| | | Max | xxx |
| Heart Rate [beats/min] | Screening | N | nn |
| | | Mean | XXX.X |
| | | SD | XXX.X |
| | | CV% | XXX.X |
| | | Min | XXX |
| | | Median | XXX.X |
| | | Max | XXX |
| Heart Rate [beats/min] | End of Study | N | nn |
| | | Mean | XXX.X |
| | | SD | XXX.X |
| | | CV% | XXX.X |
| | | Min | XXX |
| | | Median | XXX.X |
| | | Max | xxx |

Note: End of Study = Visit 9 - Day 2 - 36 hours post-dose or early termination visit for vital signs, final visit or early termination visit for body weight

Source: Listing 16.2.9.1 - Vital signs Program: Tables\k344-vs-tbl.sas



Table 14.3.5.2 - Descriptive statistics of vital signs at screening and end of study - Safety set

| Parameter | Time Point | Statistics | Safety Set<br>N=XX |
|-------------|--------------|------------|--------------------|
| W | | | |
| Weight [kg] | Screening | N | nn |
| | | Mean | XXX.X |
| | | SD | XXX.X |
| | | CV% | XXX.X |
| | | Min | XXX |
| | | Median | XXX.X |
| | | Max | xxx |
| Weight [kg] | End of Study | N | nn |
| | | Mean | XXX.X |
| | | SD | xxx.x |
| | | CV% | XXX.X |
| | | Min | XXX |
| | | Median | XXX.X |
| | | Max | XXX |

Note: End of Study = Visit 9 - Day 2 - 36 hours post-dose or early termination visit for vital signs, final visit or early termination visit for body weight

Source: Listing 16.2.9.1 - Vital signs Program: Tables\k344-vs-tbl.sas



Table 14.3.5.3 - Descriptive statistics of vital signs during the study - Safety set

| | | | | Safety | Set | |
|---|---|---|---|---|---|---|
| Parameter | Time Point | Statistics | Riluzole 50 mg<br>orodispersible film (T)<br>1 <sup>st</sup> adm.<br>N=XX | Riluzole 50 mg<br>orodispersible film (T)<br>2 <sup>nd</sup> adm.<br>N=XX | Rilutek®, 50 mg<br>riluzole tablets (R)<br>1 <sup>st</sup> adm.<br>N=XX | Rilutek®, 50 mg<br>riluzole tablets (R)<br>2 <sup>nd</sup> adm.<br>N=XX |
| Systolic Blood Pressure [mmHg] | Pre-dose | N | nn | nn | nn | nn |
| , | | Mean | XXX.X | XXX.X | XXX.X | XXX.X |
| | | SD | XXX.X | XXX.X | XXX.X | XXX.X |
| | | CV% | XXX.X | XXX.X | XXX.X | XXX.X |
| | | Min | XXX | XXX | XXX.X | XXX.X |
| | | Median | xxx.x | XXX.X | XXX.X | XXX.X |
| | | Max | XXX | XXX | XXX.X | XXX.X |
| Systolic Blood Pressure [mmHg] | 2 hours post-dose | N | nn | nn | nn | nn |
| | _ | Mean | XXX.X | XXX.X | XXX.X | XXX.X |
| | | SD | XXX.X | xxx.x | XXX.X | XXX.X |
| | | CV% | XXX.X | XXX.X | XXX.X | XXX.X |
| | | Min | XXX | XXX | XXX.X | XXX.X |
| | | Median | XXX.X | XXX.X | XXX.X | XXX.X |
| | | Max | XXX | XXX | XXX.X | XXX.X |
| Systolic Blood Pressure [mmHg] | 36 hours post-dose | N | nn | nn | nn | nn |
| | • | Mean | XXX.X | xxx.x | XXX.X | XXX.X |
| | | SD | XXX.X | XXX.X | XXX.X | XXX.X |
| | | CV% | XXX.X | XXX.X | XXX.X | XXX.X |
| | | Min | xxx | XXX | XXX.X | XXX.X |
| | | Median | XXX.X | XXX.X | XXX.X | XXX.X |
| | | Max | XXX | XXX | XXX.X | XXX.X |

Note: Subjects are summarised according to the product they actually received

Source: Listing 16.2.9.1 - Vital signs and body weight

Program: Tables\k344-vs-tbl.sas



Table 14.3.5.3 - Descriptive statistics of vital signs during the study - Safety set

| | | | | Safety | Set | |
|---|---|---|---|---|---|---|
| Parameter | Time Point | Statistics | Riluzole 50 mg<br>orodispersible film (T)<br>1 <sup>st</sup> adm.<br>N=XX | Riluzole 50 mg<br>orodispersible film (T)<br>2 <sup>nd</sup> adm.<br>N=XX | Rilutek®, 50 mg<br>riluzole tablets (R)<br>1 <sup>st</sup> adm.<br>N=XX | Rilutek®, 50 mg<br>riluzole tablets (R)<br>2 <sup>nd</sup> adm.<br>N=XX |
| Diastolic Blood Pressure [mmHg] | Pre-dose | N | nn | nn | nn | nn |
| | | Mean | XXX.X | XXX.X | XXX.X | XXX.X |
| | | SD | XXX.X | XXX.X | XXX.X | XXX.X |
| | | CV% | XXX.X | XXX.X | XXX.X | XXX.X |
| | | Min | XXX | XXX | XXX.X | XXX.X |
| | | Median | xxx.x | XXX.X | XXX.X | XXX.X |
| | | Max | XXX | XXX | XXX.X | XXX.X |
| Diastolic Blood Pressure [mmHg] | 2 hours post-dose | N | nn | nn | nn | nn |
| | • | Mean | xxx.x | XXX.X | XXX.X | XXX.X |
| | | SD | XXX.X | XXX.X | XXX.X | XXX.X |
| | | CV% | xxx.x | XXX.X | XXX.X | XXX.X |
| | | Min | XXX | XXX | XXX.X | XXX.X |
| | | Median | xxx.x | XXX.X | XXX.X | XXX.X |
| | | Max | XXX | XXX | XXX.X | XXX.X |
| Diastolic Blood Pressure [mmHg] | 36 hours post-dose | N | nn | nn | nn | nn |
| | 1 | Mean | XXX.X | XXX.X | XXX.X | XXX.X |
| | | SD | XXX.X | XXX.X | XXX.X | XXX.X |
| | | CV% | xxx.x | xxx.x | XXX.X | XXX.X |
| | | Min | XXX | XXX | XXX.X | XXX.X |
| | | Median | XXX.X | XXX.X | XXX.X | XXX.X |
| | | Max | XXX | XXX | XXX.X | XXX.X |

Note: Subjects are summarised according to the product they actually received

Source: Listing 16.2.9.1 - Vital signs and body weight

Program: Tables\k344-vs-tbl.sas



Table 14.3.5.3 - Descriptive statistics of vital signs during the study - Safety set

| | | | | Safety | Set | |
|---|---|---|---|---|---|---|
| Parameter | Time Point | Statistics | Riluzole 50 mg<br>orodispersible film (T)<br>1 <sup>st</sup> adm.<br>N=XX | Riluzole 50 mg<br>orodispersible film (T)<br>2 <sup>nd</sup> adm.<br>N=XX | Rilutek®, 50 mg<br>riluzole tablets (R)<br>1 <sup>st</sup> adm.<br>N=XX | Rilutek®, 50 mg<br>riluzole tablets (R)<br>2 <sup>nd</sup> adm.<br>N=XX |
| Heart Rate [beats/min] | Pre-dose | N | nn | nn | nn | nn |
| , | | Mean | XXX.X | XXX.X | XXX.X | XXX.X |
| | | SD | XXX.X | XXX.X | XXX.X | XXX.X |
| | | CV% | XXX.X | XXX.X | XXX.X | XXX.X |
| | | Min | XXX | XXX | XXX.X | XXX.X |
| | | Median | xxx.x | XXX.X | XXX.X | XXX.X |
| | | Max | XXX | XXX | XXX.X | XXX.X |
| Heart Rate [beats/min] | 2 hours post-dose | N | nn | nn | nn | nn |
| - | • | Mean | xxx.x | XXX.X | XXX.X | XXX.X |
| | | SD | XXX.X | XXX.X | XXX.X | XXX.X |
| | | CV% | xxx.x | XXX.X | XXX.X | XXX.X |
| | | Min | XXX | XXX | XXX.X | XXX.X |
| | | Median | xxx.x | XXX.X | XXX.X | XXX.X |
| | | Max | XXX | XXX | XXX.X | XXX.X |
| Heart Rate [beats/min] | 36 hours post-dose | N | nn | nn | nn | nn |
| | Ī | Mean | XXX.X | XXX.X | XXX.X | XXX.X |
| | | SD | XXX.X | XXX.X | XXX.X | XXX.X |
| | | CV% | XXX.X | XXX.X | XXX.X | XXX.X |
| | | Min | XXX | XXX | XXX.X | XXX.X |
| | | Median | XXX.X | XXX.X | XXX.X | XXX.X |
| | | Max | XXX | XXX | XXX.X | XXX.X |

Note: Subjects are summarised according to the product they actually received

Source: Listing 16.2.9.1 - Vital signs and body weight

Program: Tables\k344-vs-tbl.sas



Table 14.3.5.4 - Contingency tables of investigator's interpretation of mouth visual inspection during the study - Safety set

| | | Safety Set | |
|---|---|---|---|
| Time Point | Investigator's interpretation | Riluzole 50 mg<br>orodispersible film (T)<br>1 <sup>st</sup> adm.<br>N=XX | Riluzole 50 mg<br>orodispersible film (T)<br>2 <sup>nd</sup> adm.<br>N=XX |
| Pre-dose | Normal | nn (xx.x) | nn (xx.x) |
| | Abnormal, Not Clinically Significant | nn(xx.x) | nn (xx.x) |
| | Abnormal, Clinically Significant | nn(xx.x) | nn (xx.x) |
| 0.5 hour post-dose | Normal | nn(xx.x) | nn (xx.x) |
| | Abnormal, Not Clinically Significant | nn (xx.x) | nn (xx.x) |
| | Abnormal, Clinically Significant | nn(xx.x) | nn (xx.x) |
| 1 hour post-dose | Normal | nn (xx.x) | nn(xx.x) |
| | Abnormal, Not Clinically Significant | nn (xx.x) | nn (xx.x) |
| | Abnormal, Clinically Significant | nn (xx.x) | nn (xx.x) |

Note: The number and the proportion of subjects for each classification level are reported

The denominator for calculating the proportions is the number of subjects in the safety set of Riluzole 50 mg orodispersible film (T) of each administration

Source: Listing 16.2.10.3 - Mouth Visual Inspection

Program: Tables\k344-pe-tbl.sas



Table 14.3.5.5 - Descriptive statistics of dose per body weight - Safety set

| Parameter | Sex | Statistics | Safety Set<br>N=XX |
|---|---|---|---|
| Dose per body weight [mg/kg] | Females | N | nn |
| , , , , | | Mean | XXX,X |
| | | SD | XXX,X |
| | | CV% | XXX.X |
| | | Min | XXX |
| | | Median | XXX,X |
| | | Max | XXX |
| Dose per body weight [mg/kg] | Males | N | nn |
| | | Mean | XXX.X |
| | | SD | XXX.X |
| | | CV% | XXX.X |
| | | Min | XXX |
| | | Median | XXX.X |
| | | Max | XXX |
| D 1.1 11.5 // 1 | F 1 1 1 | N | |
| Dose per body weight [mg/kg] | Females and males | N | nn |
| | | Mean | XXX.X |
| | | SD | XXX.X |
| | | CV% | XXX.X |
| | | Min | XXX |
| | | Median | XXX.X |
| | | Max | XXX |

Note: The dose per body weight was calculated using the screening body weight

Source: Listing 16.2.5.2 - Dose per body weight

Program: Tables\k344-ex-tbl.sas


Table 14.3.5.6 - Descriptive statistics of wash-out - Safety set

| Parameter | Statistics | Safety Set<br>N=XX |
|---|---|---|
| Wash-out between IMP administration of Period 1 and Period 2 [days] | N | nn |
| wasii-out between him administration of Feriod Fand Feriod 2 [days] | Min | XXX |
| | Max | XXX |
| Wash-out between IMP administration of Period 2 and Period 3 [days] | N | nn |
| | Min | XXX |
| | Max | XXX |
| Wash-out between IMP administration of Period 3 and Period 4 [days] | N | nn |
| | Min | XXX |
| | Max | XXX |

Note: The wash-out is calculated as the difference in days between the dates of product administrations

Source: Listing 16.2.5.1 - Investigational medicinal products administration

Program: Tables $\k344$ -ex-tbl.sas



#### Section 16.2 - Individual Subject Data Listings Shells

| Listing 16.2.1.1 - Discontinued | subjects |
|---------------------------------|----------|
|---------------------------------|----------|

Listing 16.2.2.1 - Protocol deviations

Listing 16.2.3.1 - Subjects excluded from PK and/or safety analysis

Listing 16.2.4.1 - Subjects' disposition

Listing 16.2.4.2 - Analysis sets

Listing 16.2.4.3 - Demography

Listing 16.2.4.4 - Inclusion/Exclusion criteria not met

Listing 16.2.4.5 - Investigator's interpretation of ECG

Listing 16.2.4.6 - Tobacco consumption

Listing 16.2.5.1 - Investigational medicinal products administration

Listing 16.2.5.2 - Dose per body weight

Listing 16.2.5.3 - PK samples collection dates and times

Listing 16.2.5.4 - Riluzole concentrations (ng/mL) measured in plasma

Listing 16.2.6.1 - Riluzole plasma PK parameters

Listing 16.2.6.2 - Palatability

Listing 16.2.7.1 - Treatment-emergent adverse events

Listing 16.2.7.2 - Pre-treatment adverse events

Listing 16.2.8.1 - Individual laboratory measurements

Listing 16.2.8.2 - Investigator's interpretation of laboratory test results

Listing 16.2.9.1 - Vital signs and body weight

Listing 16.2.10.1 - Medical and surgical history

Listing 16.2.10.2 - Physical examination

Listing 16.2.10.3 - Mouth Visual Inspection

Listing 16.2.10.4 - Prior and concomitant medications

Listing 16.2.10.5 - Subjects study visits

Listing 16.2.10.6 - Fertility status and contraception

Listing 16.2.10.7 - Meals



**Listing 16.2.1.1 - Discontinued subjects** 

| Subject<br>ID | Last IMP before discontinuation | Sex | Age<br>(years) | Last<br>visit | Time elapsed from<br>last drug administration<br>(days) | Date of premature discontinuation | Primary reason for subject premature study termination |
|---|---|---|---|---|---|---|---|
| S001/001 | Riluzole 50 mg orodispersible film (T) | M | 30 | Visit 3 | 1 | ddMMMyyyy | Withdrawal by subject |
| S003/002 | Rilutek®, 50 mg riluzole tablets (R) | F | 27 | Visit 5 | 2 | ddMMMyyyy | Adverse event |
| S005/004 | Rilutek®, 50 mg riluzole tablets (R) | M | 18 | Visit 3 | 2 | ddMMMyyyy | Physician decision |
| S007/006 | Riluzole 50 mg orodispersible film (T) | F | 27 | Visit 5 | 2 | ddMMMyyyy | Adverse event |
| S011/010 | Rilutek®, 50 mg riluzole tablets (R) | M | 18 | Visit 3 | 2 | ddMMMyyyy | Physician decision |
| | | | | ••• | ••• | ••• | |

Note: Subjects are listed according to the last product they actually received before discontinuation

Program: Listings\k344-ds-lst.sas



**Listing 16.2.2.1 - Protocol deviations** 

| Subject<br>ID | Deviation<br>Number | Deviation<br>Category | | Deviation Description |
|---|---|---|---|---|
| S001/001 | 1 | Minor | Deviation from scheduled sampling time | Sample number 2 was collected outside the window of 15 min post-dose |
| S007/006 | 1 | Major | Inclusion criteria violation | Inclusion criteria violation |
| ••• | | ••• | | |

Program: Listings\k344-dv-lst.sas



Listing 16.2.3.1 - Subjects excluded from PK and/or safety analysis

| Subject<br>ID | Sex | Age<br>(years) | Enrolled<br>Set | Safety<br>Set | PK<br>Set | Reason for the exclusion |
|---|---|---|---|---|---|---|
| S010/008 | F | 30 | Y | N | N | Lack of IMP administration |
| S015/013 | F | 20 | Y | Y | N | Major protocol deviations |
| ••• | ••• | | • | • | • | |

Program: Listings\k344-ds-lst.sas



# Listing 16.2.4.1 - Subjects' disposition

| Subject<br>ID | Date of<br>Informed | Date of Screening | Date of<br>Enrolment | Date of<br>First | Date of<br>Last | Completed or | Date of Study<br>Completion or | Date of<br>End of | Reason for discontinuation |
|---|---|---|---|---|---|---|---|---|---|
| | Consent | | | Administration | Administration | Discontinued | Discontinuation | Participation | |
| S001/001 | ddMMMyyyy | ddMMMyyyy | ddMMMyyyy | ddMMMyyyy | ddMMMyyyy | Discontinued | ddMMMyyyy | ddMMMyyyy | Withdrawal by subject |
| S002/002 | ddMMMyyyy | ddMMMyyyy | ddMMMyyyy | ddMMMyyyy | ddMMMyyyy | Completed | ddMMMyyyy | ddMMMyyyy | |
| S005/003 | ddMMMyyyy | ddMMMyyyy | ddMMMyyyy | ddMMMyyyy | ddMMMyyyy | Discontinued | ddMMMyyyy | ddMMMyyyy | Adverse event |
| | | ••• | ••• | ••• | ••• | ••• | | | |

Program: Listings\k344-ds-lst.sas



## Listing 16.2.4.2 - Analysis sets

| Subject | <b>Planned Sequence</b> | Enrolled | Safety | PK | Reason for the exclusion |
|---|---|---|---|---|---|
| ID | | Set | Set | Set | |
| S001/001 | TRTR | Y | N | N | Lack of IMP intake |
| S003/002 | RTRT | Y | Y | Y | |
| ••• | | • | • | | |

Note: Subjects are listed according to the sequence they were assigned to

T: Riluzole 50 mg orodispersible film (T) R: Rilutek®, 50 mg riluzole tablets (R) Program: Listings\k344-ds-lst.sas



# Listing 16.2.4.3 - Demography

| Subject<br>ID | Sex | Race | Birth<br>Year | Age<br>(years) | Height (cm) | Body Weight (kg) | Body Mass Index (kg/m²) |
|---|---|---|---|---|---|---|---|
| S001/001 | F | White | 2001 | 20 | 170 | 55.0 | 19.0 |
| S002/002 | M | White | 1990 | 31 | 187 | 91.0 | 26.0 |
| | ••• | | | | ••• | | |

Note:Program:Listings\k344-dm-lst.sas





## Listing 16.2.4.4 - Inclusion/Exclusion criteria not met

| Subject<br>ID | Criterion | Verbatim |
|---|---|---|
| S001/001 | Inclusion criterion 4 | Body Mass Index (BMI): 18.5-29 kg/m2 inclusive |
| | ••• | <b></b> |

Program: Listings\k344-ie-lst.sas



Listing 16.2.4.5 - Investigator's interpretation of ECG

| Subject<br>ID | Time<br>Point | Assessment<br>Date/Time | Investigator's<br>Interpretation | Clinically<br>Significant<br>Abnormalites |
|---|---|---|---|---|
| S001/001 | Screening | ddMMMyyyy hh:mm | Abnormal, Not Clinically Significant | |
| S005/002 | Screening | ddMMMyyyy hh:mm | Normal | |

Program: Listings\k344-eg-lst.sas



## **Listing 16.2.4.6 - Tobacco consumption**

| Subject<br>ID | Tobacco Consumption | End of consumption Date |
|---------------|---------------------|-------------------------|
| S001/001 | Non smoker | |
| S003/003 | Ex Smoker | 2019 |

Program: Listings\k344-su-lst.sas



#### Listing 16.2.5.1 - Investigational medicinal products administration

Investigational Medicinal Product: Riluzole 50 mg orodispersible film (T)

| Subjec<br>ID | ct Adm<br>Nr. | | Administration<br>Date/time | Dissolution<br>Start<br>Time | Dissolution<br>End<br>Time | Film<br>swallowed<br>within 5<br>min? | If yes,<br>accidental<br>swallowing<br>time | Film<br>undissolved<br>at 5 min<br>after Adm.? | Fasting<br>Conditions<br>From 10 h<br>before<br>IMP Adm.? | Fasting Conditions<br>Start Date/time | Time from<br>Start of<br>Fasting<br>Conditions |
|---|---|---|---|---|---|---|---|---|---|---|---|
| S001/0 | 01 1 | Visit 3 | ddMMMyyyy hh:mm | hh:mm:ss | hh:mm:ss | N | | N | Y | ddMMMyyyy hh:mm | xx min |
| S001/0 | 01 3 | Visit 7 | ddMMMyyyy hh:mm | hh:mm:ss | hh:mm:ss | N | | N | Y | ddMMMyyyy hh:mm | xx min |
| ••• | ••• | ••• | ••• | ••• | ••• | ••• | ••• | ••• | ••• | ••• | ••• |

Note: Subjects are listed according to the product they actually received

Program: Listings\k344-ex-lst.sas



#### Listing 16.2.5.1 - Investigational medicinal products administration

Investigational Medicinal Product: Rilutek®, 50 mg riluzole tablets (R)

| | Subject<br>ID | Adm.<br>Nr. | Adm.<br>Visit | Administration<br>Date/time | Dissolution<br>Start<br>Time | Dissolution<br>End<br>Time | Film<br>swallowed<br>within 5<br>min? | If yes,<br>accidental<br>swallowing<br>time | Film<br>undissolved<br>at 5 min<br>after Adm.? | Fasting<br>Conditions<br>From 10 h<br>before<br>IMP Adm.? | Fasting Conditions<br>Start Date/time | Time from<br>Start of<br>Fasting<br>Conditions |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| • | S001/001 | 2 | Visit 5 | ddMMMyyyy hh:mm | | | | | | Y | ddMMMyyyy hh:mm | xx min |
| | S001/001 | 4 | Visit 9 | ddMMMyyyy hh:mm | | | | | | Y | ddMMMyyyy hh:mm | xx min |
| | ••• | ••• | ••• | ••• | ••• | ••• | ••• | ••• | ••• | ••• | ••• | ••• |

Note: Subjects are listed according to the product they actually received

Program: Listings\k344-ex-lst.sas



#### Listing 16.2.5.2 - Dose per body weight

Investigational Medicinal Product: Riluzole 50 mg orodispersible film (T)

| Subject<br>ID | Active<br>Ingredient | Dose<br>Administered | Body Weight at Screening | Dose per<br>Body Weight |
|---|---|---|---|---|
| | | (mg) | (kg) | (mg/kg) |
| S001/001 | Riluzole | 200 | 55.0 | 3.63 |
| ••• | ••• | ••• | | ••• |

Note: The dose per body weight is calculated using the screening body weight

Program: Listings\k344-ex-lst.sas



Listing 16.2.5.3 - PK samples collection dates and times

Investigational Medicinal Product: Riluzole 50 mg orodispersible film (T)

| Subject<br>ID | IMP Administration<br>Date/Time | IMP<br>Adm.<br>Nr. | Time Point | Sample<br>Number | Collection<br>Date/time | Time from IMP Administration |
|---|---|---|---|---|---|---|
| S001/001 | ddMMMyyyy hh:mm | 1 | Pre-dose - Within 30 min before IMP administration | 1 | ddMMMyyyy hh:mm | -xx min |
| S001/001 | ddMMMyyyy hh:mm | 1 | 15 min post-dose | 2 | ddMMMyyyy hh:mm | xx min |
| S001/001 | ddMMMyyyy hh:mm | 1 | $30 \text{ min post-dose} \pm 1 \text{ min}$ | 3 | ddMMMyyyy hh:mm | xx min |
| S001/001 | ddMMMyyyy hh:mm | 1 | 45 min post-dose $\pm 2$ min | 4 | ddMMMyyyy hh:mm | xx min |
| S001/001 | ddMMMyyyy hh:mm | 1 | 1 hour post-dose $\pm$ 3 min | 5 | ddMMMyyyy hh:mm | xx h xx min |
| S001/001 | ddMMMyyyy hh:mm | 1 | 1.25 hours post-dose $\pm$ 3 min | 6 | ddMMMyyyy hh:mm | xx h xx min |
| S001/001 | ddMMMyyyy hh:mm | 1 | 1.5 hours post-dose $\pm$ 3 min | 7 | ddMMMyyyy hh:mm | xx h xx min |
| S001/001 | ddMMMyyyy hh:mm | 1 | 2 hours post-dose $\pm$ 5 min | 8 | ddMMMyyyy hh:mm | xx h xx min |
| S001/001 | ddMMMyyyy hh:mm | 1 | 3 hours post-dose $\pm$ 5 min | 9 | ddMMMyyyy hh:mm | xx h xx min |
| S001/001 | ddMMMyyyy hh:mm | 1 | 4 hours post-dose $\pm$ 5 min | 10 | ddMMMyyyy hh:mm | xx h xx min |
| S001/001 | ddMMMyyyy hh:mm | 1 | 6 hours post-dose $\pm$ 10 min | 11 | ddMMMyyyy hh:mm | xx h xx min |
| S001/001 | ddMMMyyyy hh:mm | 1 | 8 hours post-dose $\pm$ 10 min | 12 | ddMMMyyyy hh:mm | xx h xx min |
| S001/001 | ddMMMyyyy hh:mm | 1 | 12 hours post-dose $\pm$ 10 min | 13 | ddMMMyyyy hh:mm | xx h xx min |
| S001/001 | ddMMMyyyy hh:mm | 1 | 24 hours post-dose $\pm$ 10 min | 14 | ddMMMyyyy hh:mm | xx h xx min |
| S001/001 | ddMMMyyyy hh:mm | 1 | 36 hours post-dose $\pm$ 10 min | 15 | ddMMMyyyy hh:mm | xx h xx min |
| S001/001 | ddMMMyyyy hh:mm | 3 | Pre-dose - Within 30 min before IMP administration | 31 | ddMMMyyyy hh:mm | -xx min |
| S001/001 | ddMMMyyyy hh:mm | 3 | 15 min post-dose | 32 | ddMMMyyyy hh:mm | xx min |
| S001/001 | ddMMMyyyy hh:mm | 3 | 30 min post-dose $\pm$ 1 min | 33 | ddMMMyyyy hh:mm | xx min |

Note: Subjects are listed according to the product they actually received

 $Program: Listings \backslash k344\text{-pc-lst.sas}$ 



Listing 16.2.5.3 - PK samples collection dates and times

Investigational Medicinal Product: Riluzole 50 mg orodispersible film (T)

| Subject<br>ID | IMP Administration<br>Date/Time | IMP<br>Adm.<br>Nr. | Time Point | Sample<br>Number | Collection<br>Date/time | Time from IMP Administration |
|---|---|---|---|---|---|---|
| S001/001 | ddMMMyyyy hh:mm | 3 | 45 min post-dose $\pm$ 2 min | 34 | ddMMMyyyy hh:mm | xx min |
| S001/001 | ddMMMyyyy hh:mm | 3 | 1 hour post-dose $\pm$ 3 min | 35 | ddMMMyyyy hh:mm | xx h xx min |
| S001/001 | ddMMMyyyy hh:mm | 3 | 1.25 hours post-dose $\pm$ 3 min | 36 | ddMMMyyyy hh:mm | xx h xx min |
| S001/001 | ddMMMyyyy hh:mm | 3 | 1.5 hours post-dose $\pm$ 3 min | 37 | ddMMMyyyy hh:mm | xx h xx min |
| S001/001 | ddMMMyyyy hh:mm | 3 | 2 hours post-dose $\pm$ 5 min | 38 | ddMMMyyyy hh:mm | xx h xx min |
| S001/001 | ddMMMyyyy hh:mm | 3 | 3 hours post-dose $\pm$ 5 min | 39 | ddMMMyyyy hh:mm | xx h xx min |
| S001/001 | ddMMMyyyy hh:mm | 3 | 4 hours post-dose $\pm$ 5 min | 40 | ddMMMyyyy hh:mm | xx h xx min |
| S001/001 | ddMMMyyyy hh:mm | 3 | 6 hours post-dose $\pm$ 10 min | 41 | ddMMMyyyy hh:mm | xx h xx min |
| S001/001 | ddMMMyyyy hh:mm | 3 | 8 hours post-dose $\pm$ 10 min | 42 | ddMMMyyyy hh:mm | xx h xx min |
| S001/001 | ddMMMyyyy hh:mm | 3 | $12 \text{ hours post-dose} \pm 10 \text{ min}$ | 43 | ddMMMyyyy hh:mm | xx h xx min |
| S001/001 | ddMMMyyyy hh:mm | 3 | 24 hours post-dose $\pm$ 10 min | 44 | ddMMMyyyy hh:mm | xx h xx min |
| S001/001 | ddMMMyyyy hh:mm | 3 | $36 \text{ hours post-dose} \pm 10 \text{ min}$ | 45 | ddMMMyyyy hh:mm | xx h xx min |

Note: Subjects are listed according to the product they actually received

Program: Listings\k344-pc-lst.sas



Listing 16.2.5.3 - PK samples collection dates and times

Investigational Medicinal Product: Rilutek®, 50 mg riluzole tablets (R)

| Subject<br>ID | IMP Administration<br>Date/Time | IMP<br>Adm.<br>Nr. | Time Point | Sample<br>Number | Collection<br>Date/time | Time from IMP Administration |
|---|---|---|---|---|---|---|
| S001/001 | ddMMMyyyy hh:mm | 2 | Pre-dose - Within 30 min before IMP administration | 16 | ddMMMyyyy hh:mm | -xx min |
| S001/001 | ddMMMyyyy hh:mm | 2 | 15 min post-dose | 17 | ddMMMyyyy hh:mm | xx min |
| S001/001 | ddMMMyyyy hh:mm | 2 | $30 \text{ min post-dose} \pm 1 \text{ min}$ | 18 | ddMMMyyyy hh:mm | xx min |
| S001/001 | ddMMMyyyy hh:mm | 2 | 45 min post-dose $\pm 2$ min | 19 | ddMMMyyyy hh:mm | xx min |
| S001/001 | ddMMMyyyy hh:mm | 2 | 1 hour post-dose $\pm$ 3 min | 20 | ddMMMyyyy hh:mm | xx h xx min |
| S001/001 | ddMMMyyyy hh:mm | 2 | 1.25 hours post-dose $\pm$ 3 min | 21 | ddMMMyyyy hh:mm | xx h xx min |
| S001/001 | ddMMMyyyy hh:mm | 2 | 1.5 hours post-dose $\pm$ 3 min | 22 | ddMMMyyyy hh:mm | xx h xx min |
| S001/001 | ddMMMyyyy hh:mm | 2 | 2 hours post-dose $\pm$ 5 min | 23 | ddMMMyyyy hh:mm | xx h xx min |
| S001/001 | ddMMMyyyy hh:mm | 2 | 3 hours post-dose $\pm$ 5 min | 24 | ddMMMyyyy hh:mm | xx h xx min |
| S001/001 | ddMMMyyyy hh:mm | 2 | 4 hours post-dose $\pm$ 5 min | 25 | ddMMMyyyy hh:mm | xx h xx min |
| S001/001 | ddMMMyyyy hh:mm | 2 | 6 hours post-dose $\pm$ 10 min | 26 | ddMMMyyyy hh:mm | xx h xx min |
| S001/001 | ddMMMyyyy hh:mm | 2 | 8 hours post-dose $\pm$ 10 min | 27 | ddMMMyyyy hh:mm | xx h xx min |
| S001/001 | ddMMMyyyy hh:mm | 2 | 12 hours post-dose $\pm$ 10 min | 28 | ddMMMyyyy hh:mm | xx h xx min |
| S001/001 | ddMMMyyyy hh:mm | 2 | 24 hours post-dose $\pm$ 10 min | 29 | ddMMMyyyy hh:mm | xx h xx min |
| S001/001 | ddMMMyyyy hh:mm | 2 | $36 \text{ hours post-dose} \pm 10 \text{ min}$ | 30 | ddMMMyyyy hh:mm | xx h xx min |
| S001/001 | ddMMMyyyy hh:mm | 4 | Pre-dose - Within 30 min before IMP administration | 46 | ddMMMyyyy hh:mm | -xx min |
| S001/001 | ddMMMyyyy hh:mm | 4 | 15 min post-dose | 47 | ddMMMyyyy hh:mm | xx min |
| S001/001 | ddMMMyyyy hh:mm | 4 | $30 \text{ min post-dose} \pm 1 \text{ min}$ | 48 | ddMMMyyyy hh:mm | xx min |

Note: Subjects are listed according to the product they actually received

 $Program: Listings \backslash k344\text{-pc-lst.sas}$ 



Listing 16.2.5.3 - PK samples collection dates and times

Investigational Medicinal Product: Rilutek®, 50 mg riluzole tablets (R)

| Subject<br>ID | IMP Administration<br>Date/Time | IMP<br>Adm.<br>Nr. | Time Point | Sample<br>Number | Collection<br>Date/time | Time from IMP Administration |
|---|---|---|---|---|---|---|
| S001/001 | ddMMMyyyy hh:mm | 4 | 45 min post-dose $\pm 2$ min | 49 | ddMMMyyyy hh:mm | xx min |
| S001/001 | ddMMMyyyy hh:mm | 4 | 1 hour post-dose $\pm$ 3 min | 50 | ddMMMyyyy hh:mm | xx h xx min |
| S001/001 | ddMMMyyyy hh:mm | 4 | 1.25 hours post-dose $\pm$ 3 min | 51 | ddMMMyyyy hh:mm | xx h xx min |
| S001/001 | ddMMMyyyy hh:mm | 4 | 1.5 hours post-dose $\pm$ 3 min | 52 | ddMMMyyyy hh:mm | xx h xx min |
| S001/001 | ddMMMyyyy hh:mm | 4 | 2 hours post-dose $\pm$ 5 min | 53 | ddMMMyyyy hh:mm | xx h xx min |
| S001/001 | ddMMMyyyy hh:mm | 4 | 3 hours post-dose $\pm$ 5 min | 54 | ddMMMyyyy hh:mm | xx h xx min |
| S001/001 | ddMMMyyyy hh:mm | 4 | 4 hours post-dose $\pm$ 5 min | 55 | ddMMMyyyy hh:mm | xx h xx min |
| S001/001 | ddMMMyyyy hh:mm | 4 | 6 hours post-dose $\pm$ 10 min | 56 | ddMMMyyyy hh:mm | xx h xx min |
| S001/001 | ddMMMyyyy hh:mm | 4 | 8 hours post-dose $\pm$ 10 min | 57 | ddMMMyyyy hh:mm | xx h xx min |
| S001/001 | ddMMMyyyy hh:mm | 4 | 12 hours post-dose $\pm$ 10 min | 58 | ddMMMyyyy hh:mm | xx h xx min |
| S001/001 | ddMMMyyyy hh:mm | 4 | 24 hours post-dose $\pm$ 10 min | 59 | ddMMMyyyy hh:mm | xx h xx min |
| S001/001 | ddMMMyyyy hh:mm | 4 | $36 \text{ hours post-dose} \pm 10 \text{ min}$ | 60 | ddMMMyyyy hh:mm | xx h xx min |

Note: Subjects are listed according to the product they actually received

Program: Listings\k344-pc-lst.sas



Listing 16.2.5.4 - Riluzole concentrations (ng/mL) measured in plasma

Investigational Medicinal Product: Riluzole 50 mg orodispersible film (T)

| Subject<br>ID | Period | Pre<br>dose | 0.25 h | 0.5 h | 0.75 h | 1 h | 1.25 h | 1.5 h | 2 h | 3 h | 4 h | 6 h | 8 h | 12 h | 24 h | 36 h |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| S001/001 | 1 | BLQL | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| S001/001 | 3 | BLQL | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| ••• | | | ••• | ••• | ••• | ••• | ••• | ••• | | ••• | ••• | ••• | ••• | ••• | ••• | ••• |

BLQL: Below Lower Quantification Limit (xx.xx ng/mL)

Program: pk-analysis\k344-tlf.sas



Listing 16.2.5.4 - Riluzole concentrations (ng/mL) measured in plasma

Investigational Medicinal Product: Rilutek®, 50 mg riluzole tablets (R)

| Subject<br>ID | Period | Pre<br>dose | 0.25 h | 0.5 h | 0.75 h | 1 h | 1.25 h | 1.5 h | 2 h | 3 h | 4 h | 6 h | 8 h | 12 h | 24 h | 36 h |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| S001/001 | 2 | BLQL | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| S001/001 | 4 | BLQL | xx.xx | xx.xx | XX.XX | xx.xx | xx.xx | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| ••• | | | ••• | ••• | ••• | ••• | ••• | ••• | | ••• | | ••• | ••• | ••• | ••• | ••• |

BLQL: Below Lower Quantification Limit (xx.xx ng/mL)

Program: pk-analysis\k344-tlf.sas



## Listing 16.2.6.1 - Riluzole plasma PK parameters

## Investigational Medicinal Product: Riluzole 50 mg orodispersible film (T)

| Subject | Period | Cmax | tmax | AUC <sub>0-t</sub> | AUC <sub>0-inf</sub> | <b>AUC</b> extra | <b>t</b> ½ | $\lambda_z$ | Points | $\mathbb{R}^2$ |
|---|---|---|---|---|---|---|---|---|---|---|
| ID | | (ng/mL) | (h) | (h*ng/mL) | (h*ng/mL) | (%) | (h) | (1/h) | | |
| S001/001 | 1 | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX |
| S001/001 | 3 | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | xxx.xx | XXX.XX |
| ••• | | ••• | | ••• | ••• | ••• | ••• | ••• | | ••• |

Note: Only subjects included in PK Set are listed

Program: pk-analysis\k344-tlf.sas



## Listing 16.2.6.1 - Riluzole plasma PK parameters

Investigational Medicinal Product: Rilutek®, 50 mg riluzole tablets (R)

| Subject | Period | $\mathbf{C}_{max}$ | tmax | AUC <sub>0-t</sub> | AUC <sub>0-inf</sub> | <b>AUC</b> extra | <b>t</b> ½ | $\lambda_z$ | Points | $\mathbb{R}^2$ |
|---|---|---|---|---|---|---|---|---|---|---|
| ID | | (ng/mL) | (h) | (h*ng/mL) | (h*ng/mL) | (%) | (h) | (1/h) | | |
| S001/001 | 2 | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX |
| S001/001 | 4 | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | xxx.xx | XXX.XX |
| | | | | | ••• | | | | | |

Note: Only subjects included in PK Set are listed

Program: pk-analysis\k344-tlf.sas



## Listing 16.2.6.2 - Palatability

| Subject<br>ID | IMP Administration<br>Date/Time | IMP Administration<br>Number | Time<br>Point | Assessment Date/Time | Palatability<br>Score |
|---|---|---|---|---|---|
| S001/001 | ddMMMyyyy hh:mm | 1 | Visit 3 - Day 1 - Immediately after administration | ddMMMyyyy hh:mm | 0 - Very unpleasant |
| S001/001 | ddMMMyyyy hh:mm | 3 | Visit 7 - Day 1 - Immediately after administration | ddMMMyyyy hh:mm | 1 - Unpleasant |
| | ••• | | | ••• | |

Note: Palatability has been evaluated only for Riluzole 50 mg orodispersible film (T)

Program: Listings\k344-pc-lst.sas



## Listing 16.2.7.1 - Treatment-emergent adverse events

Investigational Product: Riluzole 50 mg orodispersible film (T)

| Subject<br>ID | Adverse<br>Event<br>ID | | |
|---|---|---|---|
| 001/001 | 1 | Description: | Headache |
| | | Body Area Affected: | Head |
| | | Preferred Term <sup>1</sup> : | Headache |
| | | System Organ Class <sup>1</sup> : | Nervous system disorders |
| | | Acknowledgment Date/Time (Day) | ddMMMyyyy hh:mm (j) |
| | | Start - End Date/Time (Day): | ddMMMyyyy hh:mm (k) - ddMMMyyyy hh:mm (k+n) |
| | | Has the Adverse Event Started After the Administration of the Study Drug? | Y |
| | | Last Study Drug Administration Date/Time Before Onset | ddMMMyyyy hh:mm |
| | | Reasonable Possibility of a Causal Relationship with the Study Drug? | Y |
| | | Other Causal Relationship | |
| | | Severity: | Mild |
| | | Pattern: | Continuous |
| | | Serious? | N |
| | | Seriousness criteria: | |
| | | Action taken with Study Drug: | None |
| | | Concomitant therapy? | N |
| | | Caused Study Discontinuation? | N |
| | | Other Action Taken: | None |
| | | Outcome: | Recovered/Resolved |
| | | Comments: | |

Note: Subjects are listed according to the product they actually received

Note 1: MedDRA version 24.0 Program: Listings\k344-ae-lst.sas



## Listing 16.2.7.1 - Treatment-emergent adverse events

Investigational Product: Rilutek®, 50 mg riluzole tablets (R)

| Subject<br>ID | Adverse<br>Event<br>ID | | |
|---|---|---|---|
| 3001/001 | 2 | Description: | Headache |
| | | Body Area Affected: | Head |
| | | Preferred Term <sup>1</sup> : | Headache |
| | | System Organ Class <sup>1</sup> : | Nervous system disorders |
| | | Acknowledgment Date/Time (Day) | ddMMMyyyy hh:mm (j) |
| | | Start - End Date/Time (Day): | ddMMMyyyy hh:mm (k) - ddMMMyyyy hh:mm (k+n) |
| | | Has the Adverse Event Started After the Administration of the Study Drug? | Y |
| | | Last Study Drug Administration Date/Time Before Onset | ddMMMyyyy hh:mm |
| | | Reasonable Possibility of a Causal Relationship with the Study Drug? | Y |
| | | Other Causal Relationship | |
| | | Severity: | Mild |
| | | Pattern: | Continuous |
| | | Serious? | N |
| | | Seriousness criteria: | |
| | | Action taken with Study Drug: | None |
| | | Concomitant therapy? | N |
| | | Caused Study Discontinuation? | N |
| | | Other Action Taken: | None |
| | | Outcome: | Recovered/Resolved |
| | | Comments: | |

Note: Subjects are listed according to the product they actually received

Note 1: MedDRA version 24.0 Program: Listings\k344-ae-lst.sas



## Listing 16.2.7.2 - Pre-treatment adverse events

| Subject<br>ID | Adverse<br>Event<br>ID | | |
|---|---|---|---|
| S001/001 | 1 | Description: | Headache |
| | | Body Area Affected: | Head |
| | | Preferred Term <sup>1</sup> : | Headache |
| | | System Organ Class <sup>1</sup> : | Nervous system disorders |
| | | Acknowledgment Date/Time (Day) | ddMMMyyyy hh:mm (j) |
| | | Start - End Date/Time (Day): | ddMMMyyyy hh:mm (k) - ddMMMyyyy hh:mm (k+n) |
| | | Has the Adverse Event Started After the Administration of the Study Drug? | N |
| | | Last Study Drug Administration Date/Time Before Onset | |
| | | Reasonable Possibility of a Causal Relationship with the Study Drug? | N |
| | | Other Causal Relationship | Other, stress period |
| | | Severity: | Mild |
| | | Pattern: | Continuous |
| | | Serious? | N |
| | | Seriousness criteria: | <del></del> |
| | | Action taken with Study Drug: | None |
| | | Concomitant therapy? | N |
| | | Caused Study Discontinuation? | N |
| | | Other Action Taken: | None |
| | | Outcome: | Recovered/Resolved |
| | | Comments: | <del></del> |

Note 1: MedDRA version 24.0 Program: Listings\k344-ae-lst.sas



**Listing 16.2.8.1 - Individual laboratory measurements** 

**Category of Laboratory Parameters: BLOOD CHEMISTRY** 

| Subject<br>ID | Time<br>Point | Collection<br>Date/time | Parameter | Value and<br>Abnormality <sup>1</sup> | Normal Range or<br>Reference Value | Clinically Significant? |
|---|---|---|---|---|---|---|
| S001/001 | Screening | ddMMMyyyy hh:mm | Sodium [mmol/L] | 138 [N] | 136 - 145 | N |
| S001/001 | Screening | ddMMMyyyy hh:mm | Potassium [mmol/L] | 4.4 [N] | 3.5 - 5.1 | N |
| S001/001 | Screening | ddMMMyyyy hh:mm | Calcium [mmol/L] | 2.27 [N] | 2.10 - 2.55 | N |
| S001/001 | Screening | ddMMMyyyy hh:mm | Chloride [mmol/L] | 103 [N] | 96 - 110 | N |
| S001/001 | Screening | ddMMMyyyy hh:mm | Phosphate [mmol/L] | 0.84 [L] | 0.87 - 1.45 | N |
| S001/001 | Screening | ddMMMyyyy hh:mm | Alkaline Phosphatase [U/L] | 95 [N] | <= 129 | N |
| S001/001 | Screening | ddMMMyyyy hh:mm | Gamma Glutamyl Transferase [U/L] | 17 [N] | <= 66 | N |
| S001/001 | Screening | ddMMMyyyy hh:mm | Aspartate Aminotransferase [U/L] | 24 [N] | <= 50 | N |
| S001/001 | Screening | ddMMMyyyy hh:mm | Alanine Aminotransferase [U/L] | 30 [N] | <= 50 | N |
| ••• | ••• | ••• | | ••• | | |
| S001/001 | End of Study | ddMMMyyyy hh:mm | Sodium [mmol/L] | 138 [N] | 136 - 145 | N |
| S001/001 | End of Study | ddMMMyyyy hh:mm | Potassium [mmol/L] | 4.4 [N] | 3.5 - 5.1 | N |
| S001/001 | End of Study | ddMMMyyyy hh:mm | Calcium [mmol/L] | 2.27 [N] | 2.10 - 2.55 | N |
| S001/001 | End of Study | ddMMMyyyy hh:mm | Chloride [mmol/L] | 103 [N] | 96 - 110 | N |
| S001/001 | End of Study | ddMMMyyyy hh:mm | Phosphate [mmol/L] | 0.84 [L] | 0.87 - 1.45 | N |
| S001/001 | End of Study | ddMMMyyyy hh:mm | Alkaline Phosphatase [U/L] | 95 [N] | <= 129 | N |
| S001/001 | End of Study | ddMMMyyyy hh:mm | Gamma Glutamyl Transferase [U/L] | 17 [N] | <= 66 | N |
| S001/001 | End of Study | ddMMMyyyy hh:mm | Aspartate Aminotransferase [U/L] | 24 [N] | <= 50 | N |
| S001/001 | End of Study | ddMMMyyyy hh:mm | Alanine Aminotransferase [U/L] | 30 [N] | <= 50 | N |

Note 1: N=Normal, H=Higher than upper normal limit, L=Lower than lower normal limit

 $Program: Listings \verb|\k344-lb-lst.sas|$ 



**Listing 16.2.8.1 - Individual laboratory measurements** 

**Category of Laboratory Parameters: HEMATOLOGY** 

| Subject<br>ID | Time<br>Point | Collection<br>Date/time | Parameter | Value and Abnormality <sup>1</sup> | Normal Range or<br>Reference Value | Clinically<br>Significant? |
|---|---|---|---|---|---|---|
| S001/001 | Screening | ddMMMyyyy hh:mm | Leukocytes [10^9/L] | 10.02 [H] | 4.00 - 10.00 | N |
| S001/001 | Screening | ddMMMyyyy hh:mm | Erythrocytes [10^12/L] | 5.19 [N] | 4.30 - 5.90 | N |
| S001/001 | Screening | ddMMMyyyy hh:mm | Hemoglobin [g/dL] | 15.4 [N] | 14.0 - 18.0 | N |
| S001/001 | Screening | ddMMMyyyy hh:mm | Hemoglobin [mmol/L] | 9.6 [N] | 8.7 - 11.2 | N |
| S001/001 | Screening | ddMMMyyyy hh:mm | Hematocrit [%] | 44 [N] | 42 - 52 | N |
| S001/001 | Screening | ddMMMyyyy hh:mm | Ery. Mean Corpuscular Volume [fL] | 84 [N] | 83 - 100 | N |
| S001/001 | Screening | ddMMMyyyy hh:mm | Ery. Mean Corpuscular Hemoglobin [pg] | 30 [N] | 27 - 34 | N |
| S001/001 | Screening | ddMMMyyyy hh:mm | Ery. Mean Corpuscular HGB Concentration [g/dL] | 35 [N] | 32 - 36 | N |
| | | | <b></b> | | | |
| S001/001 | End of Study | ddMMMyyyy hh:mm | Leukocytes [10^9/L] | 10.02 [H] | 4.00 - 10.00 | N |
| S001/001 | End of Study | ddMMMyyyy hh:mm | Erythrocytes [10^12/L] | 5.19 [N] | 4.30 - 5.90 | N |
| S001/001 | End of Study | ddMMMyyyy hh:mm | Hemoglobin [g/dL] | 15.4 [N] | 14.0 - 18.0 | N |
| S001/001 | End of Study | ddMMMyyyy hh:mm | Hemoglobin [mmol/L] | 9.6 [N] | 8.7 - 11.2 | N |
| S001/001 | End of Study | ddMMMyyyy hh:mm | Hematocrit [%] | 44 [N] | 42 - 52 | N |
| S001/001 | End of Study | ddMMMyyyy hh:mm | Ery. Mean Corpuscular Volume [fL] | 84 [N] | 83 - 100 | N |
| S001/001 | End of Study | ddMMMyyyy hh:mm | Ery. Mean Corpuscular Hemoglobin [pg] | 30 [N] | 27 - 34 | N |
| S001/001 | End of Study | ddMMMyyyy hh:mm | Ery. Mean Corpuscular HGB Concentration [g/dL] | 35 [N] | 32 - 36 | N |

Note 1: N=Normal, H=Higher than upper normal limit, L=Lower than lower normal limit

Program: Listings\k344-lb-lst.sas



## **Listing 16.2.8.1 - Individual laboratory measurements**

**Category of Laboratory Parameters: COTININE** 

| Subject<br>ID | Time<br>Point | Collection<br>Date/time | Parameter | Value and Abnormality <sup>1</sup> | Normal Range or<br>Reference Value | Clinically Significant? |
|---|---|---|---|---|---|---|
| S001/001 | Screening | ddMMMyyyy hh:mm | Cotinine | Negative [N] | Negative | N |
| ••• | ••• | ••• | ••• | ••• | ••• | ••• |

Note 1: N=Normal, A=Different from reference value

Program: Listings\k344-lb-lst.sas



**Listing 16.2.8.1 - Individual laboratory measurements** 

**Category of Laboratory Parameters: URINE ANALYSIS** 

| Subject<br>ID | Time<br>Point | Collection<br>Date/time | Parameter | Value and<br>Abnormality <sup>1</sup> | Normal Range or<br>Reference Value | Clinically<br>Significant? |
|---|---|---|---|---|---|---|
| S001/001 | Screening | ddMMMyyyy hh:mm | Urobilinogen | Normal [N] | Normal | N |
| S001/001 | Screening | ddMMMyyyy hh:mm | Urinary Bilirubin | Absent [N] | Absent | N |
| S001/001 | Screening | ddMMMyyyy hh:mm | Ketones | Absent [N] | Absent | N |
| S001/001 | Screening | ddMMMyyyy hh:mm | Urinary Hemoglobin | +++ [A] | Absent | N |
| S001/001 | Screening | ddMMMyyyy hh:mm | Urinary Leukocytes | Absent [N] | Absent | N |
| S001/001 | Screening | ddMMMyyyy hh:mm | Sediment Examination | Checked | | |
| S001/001 | Screening | ddMMMyyyy hh:mm | Urinary Sediment Leukocytes | Absent [N] | Absent or 0-2 per field | N |
| S001/001 | Screening | ddMMMyyyy hh:mm | Urinary Sediment Erythrocytes | 0-2 per field [N] | Absent or 0-2 per field | N |
| | | ••• | | | ••• | |
| S001/001 | End of Study | ddMMMyyyy hh:mm | Urobilinogen | Normal [N] | Normal | N |
| S001/001 | End of Study | ddMMMyyyy hh:mm | Urinary Bilirubin | Absent [N] | Absent | N |
| S001/001 | End of Study | ddMMMyyyy hh:mm | Ketones | Absent [N] | Absent | N |
| S001/001 | End of Study | ddMMMyyyy hh:mm | Urinary Hemoglobin | +++ [A] | Absent | N |
| S001/001 | End of Study | ddMMMyyyy hh:mm | Urinary Leukocytes | Absent [N] | Absent | N |
| S001/001 | End of Study | ddMMMyyyy hh:mm | Sediment Examination | Checked | | |
| S001/001 | End of Study | ddMMMyyyy hh:mm | Urinary Sediment Leukocytes | Absent [N] | Absent or 0-2 per field | N |
| S001/001 | End of Study | ddMMMyyyy hh:mm | Urinary Sediment Erythrocytes | 0-2 per field [N] | Absent or 0-2 per field | N |

Note 1: N=Normal, A=Different from reference value

Program: Listings\k344-lb-lst.sas



**Listing 16.2.8.1 - Individual laboratory measurements** 

# **Category of Laboratory Parameters: URINE DRUG SCREENING**

| Subject<br>ID | Time<br>Point | Collection<br>Date/time | Parameter | Value and<br>Abnormality <sup>1</sup> | Normal Range or<br>Reference Value | Clinically Significant? |
|---|---|---|---|---|---|---|
| S001/001 | Screening | ddMMMyyyy hh:mm | Amphetamine | Negative [N] | Negative | N |
| S001/001 | Screening | ddMMMyyyy hh:mm | Cannabinoids | Negative [N] | Negative | N |
| S001/001 | Screening | ddMMMyyyy hh:mm | Cocaine | Negative [N] | Negative | N |
| S001/001 | Screening | ddMMMyyyy hh:mm | Ecstasy | Negative [N] | Negative | N |
| S001/001 | Screening | ddMMMyyyy hh:mm | Methamphetamine | Negative [N] | Negative | N |
| S001/001 | Screening | ddMMMyyyy hh:mm | Opiate | Negative [N] | Negative | N |

Note 1: N=Normal, A=Different from reference value

Program: Listings\k344-lb-lst.sas



#### **Listing 16.2.8.1 - Individual laboratory measurements**

**Category of Laboratory Parameters: VIROLOGY** 

| Subject<br>ID | Time<br>Point | Collection<br>Date/time | Parameter | Value and Abnormality <sup>1</sup> | Normal Range or<br>Reference Value | Clinically Significant? |
|---|---|---|---|---|---|---|
| S001/001 | Screening | ddMMMyyyy hh:mm | Hepatitis B Virus Surface Antigen | Negative [N] | Negative | N |
| S001/001 | Screening | ddMMMyyyy hh:mm | Hepatitis C Virus Antibody | Negative [N] | Negative | N |
| S001/001 | Screening | ddMMMyyyy hh:mm | HIV Ag/Ab Combo | Negative [N] | Negative | N |
| ••• | | ••• | | ••• | ••• | ••• |

Note 1: N=Normal, A=Different from reference value \_

Program: Listings\k344-lb-lst.sas



#### **Listing 16.2.8.1 - Individual laboratory measurements**

# Category of Laboratory Parameters: ALCOHOL BREATH TEST AND PREGNANCY TEST

| Subject<br>ID | Time<br>Point | Collection Date/time | Parameter | Value and<br>Abnormality <sup>1</sup> | Normal Range or<br>Reference Value | Clinically Significant? |
|---|---|---|---|---|---|---|
| S001/001 | Screening | ddMMMyyyy hh:mm | Pregnancy Test | Negative [N] | Negative | N |
| S001/001 | Visit 2 - Day -1 | ddMMMyyyy hh:mm | Pregnancy Test | Negative [N] | Negative | N |
| S001/001 | Visit 2 - Day -1 | ddMMMyyyy hh:mm | Alcohol Breath Test | Negative [N] | Negative | N |
| | ••• | ••• | <b></b> | | ••• | |

Note 1: N=Normal, A=Different from reference value

Program: Listings\k344-lb-lst.sas



Listing 16.2.8.2 - Investigator's interpretation of laboratory test results

| Subject<br>ID | Time<br>Point | Assessment<br>Date | Investigator's<br>Interpretation | Clinically<br>Significant<br>Abnormalites |
|---|---|---|---|---|
| S001/001 | Screening | ddMMMyyyy | Abnormal, Not Clinically Significant | |
| S001/001 | End of Study | ddMMMyyyy | Abnormal, Not Clinically Significant | |

Program: Listings\k344-lb-lst.sas



Listing 16.2.9.1 - Vital signs and body weight

| Subject<br>ID | Time<br>Point | Assessment<br>Date/Time | Parameter | Value and<br>Abnormality <sup>1</sup> | Normal<br>Range | Clinically Significant? |
|---|---|---|---|---|---|---|
| S001/001 | Screening | ddMMMyyyy hh:mm | Systolic Blood Pressure [mmHg] | 96 [L] | 100-139 | N |
| S001/001 | Screening | ddMMMyyyy hh:mm | Diastolic Blood Pressure [mmHg] | 58 [N] | 50-89 | N |
| S001/001 | Screening | ddMMMyyyy hh:mm | Heart Rate [beats/min] | 88 [N] | 50-90 | N |
| S001/001 | Screening | ddMMMyyyy hh:mm | Weight [kg] | 55.5 | | N |
| S001/001 | Visit 3 - Pre-dose | ddMMMyyyy hh:mm | Systolic Blood Pressure [mmHg] | 96 [L] | 100-139 | N |
| S001/001 | Visit 3 - Pre-dose | ddMMMyyyy hh:mm | Diastolic Blood Pressure [mmHg] | 58 [N] | 50-89 | N |
| S001/001 | Visit 3 - Pre-dose | ddMMMyyyy hh:mm | Heart Rate [beats/min] | 88 [N] | 50-90 | N |
| S001/001 | Visit 3 - 2 hours post-dose | ddMMMyyyy hh:mm | Systolic Blood Pressure [mmHg] | 96 [L] | 100-139 | N |
| S001/001 | Visit 3 - 2 hours post-dose | ddMMMyyyy hh:mm | Diastolic Blood Pressure [mmHg] | 58 [N] | 50-89 | N |
| S001/001 | Visit 3 - 2 hours post-dose | ddMMMyyyy hh:mm | Heart Rate [beats/min] | 88 [N] | 50-90 | N |
| S001/001 | Visit 3 - 36 hours post-dose | ddMMMyyyy hh:mm | Systolic Blood Pressure [mmHg] | 96 [L] | 100-139 | N |
| S001/001 | Visit 3 - 36 hours post-dose | ddMMMyyyy hh:mm | Diastolic Blood Pressure [mmHg] | 58 [N] | 50-89 | N |
| S001/001 | Visit 3 - 36 hours post-dose | ddMMMyyyy hh:mm | Heart Rate [beats/min] | 88 [N] | 50-90 | N |
| S001/001 | Visit 5 - Pre-dose | ddMMMyyyy hh:mm | Systolic Blood Pressure [mmHg] | 96 [L] | 100-139 | N |
| S001/001 | Visit 5 - Pre-dose | ddMMMyyyy hh:mm | Diastolic Blood Pressure [mmHg] | 58 [N] | 50-89 | N |
| S001/001 | Visit 5 - Pre-dose | ddMMMyyyy hh:mm | Heart Rate [beats/min] | 88 [N] | 50-90 | N |
| S001/001 | Visit 5 - 2 hours post-dose | ddMMMyyyy hh:mm | Systolic Blood Pressure [mmHg] | 96 [L] | 100-139 | N |
| S001/001 | Visit 5 - 2 hours post-dose | ddMMMyyyy hh:mm | Diastolic Blood Pressure [mmHg] | 58 [N] | 50-89 | N |
| S001/001 | Visit 5 - 2 hours post-dose | ddMMMyyyy hh:mm | Heart Rate [beats/min] | 88 [N] | 50-90 | N |
| S001/001 | Visit 5 - 36 hours post-dose | ddMMMyyyy hh:mm | Systolic Blood Pressure [mmHg] | 96 [L] | 100-139 | N |
| S001/001 | Visit 5 - 36 hours post-dose | ddMMMyyyy hh:mm | Diastolic Blood Pressure [mmHg] | 58 [N] | 50-89 | N |
| S001/001 | Visit 5 - 36 hours post-dose | ddMMMyyyy hh:mm | Heart Rate [beats/min] | 88 [N] | 50-90 | N |
| S001/001 | Visit 7 - Pre-dose | ddMMMyyyy hh:mm | Systolic Blood Pressure [mmHg] | 96 [L] | 100-139 | N |
| S001/001 | Visit 7 - Pre-dose | ddMMMyyyy hh:mm | Diastolic Blood Pressure [mmHg] | 58 [N] | 50-89 | N |
| S001/001 | Visit 7 - Pre-dose | ddMMMyyyy hh:mm | Heart Rate [beats/min] | 88 [N] | 50-90 | N |

Note 1: N=Normal, H=Higher than upper normal limit, L=Lower than lower normal limit

Program: Listings\k344-vs-lst.sas



Listing 16.2.9.1 - Vital signs and body weight

| Subject<br>ID | Time<br>Point | Assessment<br>Date/Time | Parameter | Value and Abnormality <sup>1</sup> | Normal<br>Range | Clinically Significant? |
|---|---|---|---|---|---|---|
| S001/001 | Visit 7 - 2 hours post-dose | ddMMMyyyy hh:mm | Systolic Blood Pressure [mmHg] | 96 [L] | 100-139 | N |
| S001/001 | Visit 7 - 2 hours post-dose | ddMMMyyyy hh:mm | Diastolic Blood Pressure [mmHg] | 58 [N] | 50-89 | N |
| S001/001 | Visit 7 - 2 hours post-dose | ddMMMyyyy hh:mm | Heart Rate [beats/min] | 88 [N] | 50-90 | N |
| S001/001 | Visit 7 - 36 hours post-dose | ddMMMyyyy hh:mm | Systolic Blood Pressure [mmHg] | 96 [L] | 100-139 | N |
| S001/001 | Visit 7 - 36 hours post-dose | ddMMMyyyy hh:mm | Diastolic Blood Pressure [mmHg] | 58 [N] | 50-89 | N |
| S001/001 | Visit 7 - 36 hours post-dose | ddMMMyyyy hh:mm | Heart Rate [beats/min] | 88 [N] | 50-90 | N |
| S001/001 | Visit 9 - Pre-dose | ddMMMyyyy hh:mm | Systolic Blood Pressure [mmHg] | 96 [L] | 100-139 | N |
| S001/001 | Visit 9 - Pre-dose | ddMMMyyyy hh:mm | Diastolic Blood Pressure [mmHg] | 58 [N] | 50-89 | N |
| S001/001 | Visit 9 - Pre-dose | ddMMMyyyy hh:mm | Heart Rate [beats/min] | 88 [N] | 50-90 | N |
| S001/001 | Visit 9 - 2 hours post-dose | ddMMMyyyy hh:mm | Systolic Blood Pressure [mmHg] | 96 [L] | 100-139 | N |
| S001/001 | Visit 9 - 2 hours post-dose | ddMMMyyyy hh:mm | Diastolic Blood Pressure [mmHg] | 58 [N] | 50-89 | N |
| S001/001 | Visit 9 - 2 hours post-dose | ddMMMyyyy hh:mm | Heart Rate [beats/min] | 88 [N] | 50-90 | N |
| S001/001 | Visit 9 - 36 hours post-dose | ddMMMyyyy hh:mm | Systolic Blood Pressure [mmHg] | 96 [L] | 100-139 | N |
| S001/001 | Visit 9 - 36 hours post-dose | ddMMMyyyy hh:mm | Diastolic Blood Pressure [mmHg] | 58 [N] | 50-89 | N |
| S001/001 | Visit 9 - 36 hours post-dose | ddMMMyyyy hh:mm | Heart Rate [beats/min] | 88 [N] | 50-90 | N |
| S001/001 | End of Study | ddMMMyyyy hh:mm | Weight [kg] | 55.5 | | N |
| | | | | | | ••• |

Note 1: N=Normal, H=Higher than upper normal limit, L=Lower than lower normal limit

Program: Listings\k344-vs-lst.sas



# Listing 16.2.10.1 - Medical and surgical history

| Subject<br>ID | Category | Disease/Surgery<br>ID | | |
|---|---|---|---|---|
| S001/001 | Medical History | M1 | Verbatim: | Left shoulder luxation |
| | | | Preferred Term 1: | Joint dislocation |
| | | | System Organ Class 1: | Injury, poisoning and procedural complications |
| | | | Disease Start - End Date: | 2012 - 2012 |
| | Surgery | S1 | Verbatim: | Right knee meniscectomy |
| | | | Preferred Term 1: | Meniscus removal |
| | | | System Organ Class 1: | Surgical and medical procedures |
| | | | Surgery Date: | 04NOV1980 |
| | ••• | ••• | | |

Note 1: MedDRA version 24.0 Program: Listings\k344-mh-lst.sas



# Listing 16.2.10.2 - Physical examination

| Subject<br>ID | Time Point | Physical<br>Examination<br>Date | | |
|---|---|---|---|---|
| S001/001 | Screening | ddMMMyyyy | Investigator's Interpretation | Normal |
| | End of Study | ddMMMyyyy | Investigator's Interpretation: | Abnormal, Clinically Significant |
| | | | Clinically Significant Abnormalities: | Left shoulder luxation |
| | | | Preferred Term <sup>1</sup> : | Joint dislocation |
| | | | System Organ Class 1: | Injury, poisoning and procedural complications |
| | ••• | ••• | | <b></b> |

Note 1: MedDRA version 24.0 Program: Listings\k344-pe-lst.sas



#### **Listing 16.2.10.3 - Mouth Visual Inspection**

| Subject<br>ID | Time Point | Physical<br>Examination<br>Date | | |
|---|---|---|---|---|
| S001/001 | Visit 3 - Pre-dose | ddMMMyyyy | Investigator's Interpretation | Normal |
| S001/001 | Visit 3 - 0.5 hour post-dose | ddMMMyyyy | Investigator's Interpretation | Abnormal, Not Clinically Significant |
| S001/001 | Visit 3 - 1 hour post-dose | ddMMMyyyy | Investigator's Interpretation:<br>Clinically Significant Abnormalities:<br>Preferred Term <sup>1</sup> :<br>System Organ Class <sup>1</sup> : | Abnormal, Clinically Significant Left shoulder luxation Joint dislocation Injury, poisoning and procedural complications |
| S001/001 | Visit 7 - Pre-dose | ddMMMyyyy | Investigator's Interpretation | Normal |
| S001/001 | Visit 7 - 0.5 hour post-dose | ddMMMyyyy | Investigator's Interpretation | Abnormal, Not Clinically Significant |
| S001/001 | Visit 7 - 1 hour post-dose | ddMMMyyyy | Investigator's Interpretation:<br>Clinically Significant Abnormalities:<br>Preferred Term <sup>1</sup> :<br>System Organ Class <sup>1</sup> : | Abnormal, Clinically Significant Left shoulder luxation Joint dislocation Injury, poisoning and procedural complications |

Note: Mouth visual inspection has been evaluated only for Riluzole 50 mg orodispersible film (T)

Note 1: MedDRA version 24.0 Program: Listings\k344-pe-lst.sas



Listing 16.2.10.4 - Prior and concomitant medications

| Subject<br>ID | Category | Medication<br>ID | | |
|---|---|---|---|---|
| S001/001 | Prior | 1 | Verbatim: | Alerid |
| | | | Standardised Medication Name 1: | Alerid |
| | | | Active Ingredients 1: | Cetirizine hydrochloride |
| | | | Medication Class 1, 2: | Piperazine derivatives (R06AE) |
| | | | Indication: | Pollinosis |
| | | | Dose: | 10 mg |
| | | | Start - End Date/Time: | 2013 - Ongoing |
| | | | Frequency - Dosage Form - Route: | 1 time per day - Tablet - Oral |
| | | | Related to: | Disease M1 |
| | Concomitant | 2 | Verbatim: | Paracen |
| | | | Standardised Medication Name 1: | Paracen |
| | | | Active Ingredients 1: | Paracetamol |
| | | | Medication Class <sup>1, 2</sup> : | Anilides (N02BE) |
| | | | Indication: | Headache |
| | | | Dose: | 500 mg |
| | | | Start - End Date/Time: | 15JUN2016 19:08 - 15JUN2016 19:08 |
| | | | Frequency - Dosage Form - Route: | Once - Tablet - Oral |
| | | | Related to: | Adverse Event 1 |
| | | | | <b></b> |

Note 1: WHO Drug Dictionary Enhanced March 1, 2021

Note 2: Anatomical Therapeutic Chemical classification, 4th level term

Program: Listings\k344-cm-lst.sas



Listing 16.2.10.5 - Subjects study visits

| Subject<br>ID | Visit | Visit Start Date (Day) | Visit End Date (Day) | Home discharge<br>Date/time |
|---|---|---|---|---|
| S001/001 | Visit 1 - Screening - Day -14/-2 | ddMMMyyyy (-j) | | |
| S001/001 | Period 1 - Visit 2 - Day -1 | ddMMMyyyy (-1) | <del></del> | |
| S001/001 | Period 1 - Visit 3 - Days 1-2 | ddMMMyyyy (1) | ddMMMyyyy (2) | ddMMMyyyy (2) hh:mm |
| S001/001 | Period 1 - Visit 4 - Day -1 | ddMMMyyyy (k-1) | | |
| S001/001 | Period 2 - Visit 5 - Days 1-2 | ddMMMyyyy (k) | ddMMMyyyy (k+1) | ddMMMyyyy (k+1) hh:mm |
| S001/001 | Period 1 - Visit 6 - Day -1 | ddMMMyyyy (n-1) | | |
| S001/001 | Period 2 - Visit 7 - Days 1-2 | ddMMMyyyy (n) | ddMMMyyyy (n+1) | ddMMMyyyy (n+1) hh:mm |
| S001/001 | Period 1 - Visit 8 - Day -1 | ddMMMyyyy (p-1) | | |
| S001/001 | Period 2 - Visit 9 - Days 1-2 | ddMMMyyyy (p) | ddMMMyyyy (p+1) | |
| S001/001 | Final Visit | ddMMMyyyy (p+1) | <del></del> | ddMMMyyyy (p+1) hh:mm |
| | | | <b></b> | |

Program: Listings\k344-sv-lst.sas





## Listing 16.2.10.6 - Fertility status and contraception

| Subject<br>ID | Chilbearing Potential? | Non-childbearing<br>Potential<br>Status Onset | Menopausal<br>Status? | Date of<br>Menopause | Surgical<br>Sterilisation? | Surgical<br>Sterilisation<br>Date | Reliable<br>Contraceptive<br>Method Used? |
|---|---|---|---|---|---|---|---|
| S001/001 | No | ddMMMyyyy | Yes | MMMyyyy | Yes | ddMMMyyyy | |
| ••• | | ••• | ••• | ••• | ••• | ••• | ••• |

Note: Only female subjects are listed Program: Listings\k344-rp-lst.sas



**Listing 16.2.10.7 - Meals** 

Investigational Medicinal Product: Riluzole 50 mg orodispersible film (T)

| Subject<br>ID | IMP<br>Administration<br>Date/Time | Meal<br>Nr | Standardised<br>Meal | Time Point | Meal<br>Served? | Meal Start<br>Date/time | Elapsed<br>Time |
|---|---|---|---|---|---|---|---|
| S001/001 | ddMMMyyyy hh:mm | 1 | Lunch | Visit 3 - Day 1 –5 hours post-dose | Y | ddMMMyyyy hh:mm | xx h xx min |
| S001/001 | ddMMMyyyy hh:mm | 2 | Dinner | Visit 3 - Day 1 −12 hours post-dose | Y | ddMMMyyyy hh:mm | xx h xx min |
| S001/001 | | 3 | Breakfast | Visit 3 - Day 2 - at about 08:00 | Y | ddMMMyyyy hh:mm | |
| S001/001 | | 4 | Lunch | Visit 3 - Day 2 - at about 13:00 | Y | ddMMMyyyy hh:mm | |
| S001/001 | ddMMMyyyy hh:mm | 9 | Lunch | Visit 7 - Day 1 –5 hours post-dose | Y | ddMMMyyyy hh:mm | xx h xx min |
| S001/001 | ddMMMyyyy hh:mm | 10 | Dinner | Visit 7 - Day 1 –12 hours post-dose | Y | ddMMMyyyy hh:mm | xx h xx min |
| S001/001 | | 11 | Breakfast | Visit 7 - Day 2 -at about 08:00 | Y | ddMMMyyyy hh:mm | |
| S001/001 | | 12 | Lunch | Visit 7 - Day 2 - at about 13:00 | Y | ddMMMyyyy hh:mm | |
| ••• | ••• | | | | ••• | ••• | ••• |

Note: Subjects are listed according to the product they actually received

Program: Listings\k344-ml-lst.sas



**Listing 16.2.10.7 - Meals** 

Investigational Medicinal Product: Rilutek®, 50 mg riluzole tablets (R)

| Subject<br>ID | IMP<br>Administration<br>Date/Time | Meal<br>Nr | Standardised<br>Meal | Time Point | Meal<br>Served? | Meal Start<br>Date/time | Elapsed<br>Time |
|---|---|---|---|---|---|---|---|
| S001/001 | ddMMMyyyy hh:mm | 5 | Lunch | Visit 5 - Day 1 –5 hours post-dose | Y | ddMMMyyyy hh:mm | xx h xx min |
| S001/001 | ddMMMyyyy hh:mm | 6 | Dinner | Visit 5 - Day 1 –12 hours post-dose | Y | ddMMMyyyy hh:mm | xx h xx min |
| S001/001 | | 7 | Breakfast | Visit 5 - Day 2 -at about 08:00 | Y | ddMMMyyyy hh:mm | |
| S001/001 | | 8 | Lunch | Visit 5 - Day 2 - at about 13:00 | Y | ddMMMyyyy hh:mm | |
| S001/001 | ddMMMyyyy hh:mm | 13 | Lunch | Visit 9 - Day 1 –5 hours post-dose | Y | ddMMMyyyy hh:mm | xx h xx min |
| S001/001 | ddMMMyyyy hh:mm | 14 | Dinner | Visit 9 - Day 1 −12 hours post-dose | Y | ddMMMyyyy hh:mm | xx h xx min |
| S001/001 | | 15 | Breakfast | Visit 9 - Day 2 – at about 08:00 | Y | ddMMMyyyy hh:mm | |
| S001/001 | | 16 | Lunch | Visit 9 - Day 2 - at about 13:00 | Y | ddMMMyyyy hh:mm | |

Note: Subjects are listed according to the product they actually received

Program: Listings\k344-ml-lst.sas